

A Randomised, Phase 1b, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacokinetics, and Antiviral Activity Of RV299 Against Respiratory Syncytial Virus in the Viral Challenge Model

Protocol No: REVD002

hVIVO Study No: VIR-CST-001

CCI

For: hVIVO Services Ltd

# **CONTENTS**

| 1. | STATISTICAL ANALYSIS PLAN APPROVAL FORM | 5 |
|---|---|---|
| 2. | STATISTICAL ANALYSIS PLAN AUTHOR | 6 |
| 3. | LIST OF ABBREVIATIONS | 7 |
| 4. | INTRODUCTION | 9 |
| 5. | STUDY OBJECTIVES | 10 |
| | 5.1. Primary Objective | 10 |
| | 5.2. Secondary Objectives | 10 |
| 6. | STUDY DESIGN | 11 |
| 0. | 6.1. Summary of Study Design | |
| | 6.2. Randomisation / Treatment Allocation and Blinding | |
| | 6.3. Time and Events Schedule | |
| | 6.4. Interim Analysis / Data Monitoring | |
| 7. | STUDY ENDPOINTS | 20 |
| | 7.1. Primary Endpoint | 20 |
| | 7.2. Secondary Endpoints | 20 |
| | CCI | |
| CCI | | |
| 9. | STUDY POPULATIONS | 24 |
| | 9.1. Intent-to-Treat (ITT) Population | 24 |
| | 9.2. Intent-to-Treat Infected (ITT-I) Population | 24 |
| | 9.3. Intent-to-Treat Infected Analysis Population A (ITT-A) Population | 24 |
| | 9.4. Intent-to-Treat Infected Analysis Population B (ITT-B) Population | 25 |
| | 9.5. Per Protocol (PP) Population | 25 |
| | 9.6. Safety Population | 25 |
| | 9.7. PK Population | 25 |
| 10. | PLANNED STATISTICAL METHODS | 26 |
| | 10.1. Statistical Considerations | 26 |
| | 10.1.1. General Definitions | 26 |
| | 10.1.2. Data Presentation | 26 |
| | 10.1.3. Early Withdrawal Visit | 28 |

| | 10.1.4. Statistical Testing and Estimation | 28 |
|---|---|---|
| | 10.1.5. Handling of Dropouts or Missing Data | 28 |
| | 10.1.6. Interim Analysis and Data Monitoring | 29 |
| | 10.1.7. Multiple Comparison/Multiplicity | 29 |
| | 10.1.8. Model Checking and Sensitivity Analyses | 29 |
| | 10.1.9. Data Conversion (CDISC) | 29 |
| | 10.1.10. Software | 29 |
| | 10.2. Participant Disposition | 29 |
| | 10.3. Protocol Deviations | 29 |
| | 10.4. Demographic and Other Baseline Characteristics | 30 |
| | 10.4.1. Demographics | 30 |
| | 10.4.2. Substance Use History and Recreational Drugs of Misuse | 30 |
| | 10.4.3. Reproductive Status and Contraceptive Use | 30 |
| | 10.4.4. Medical History | 30 |
| | 10.5. Prior and Concomitant Medications | 30 |
| | 10.6. IMP Exposure and Compliance | 31 |
| | 10.7. Statistical Analysis | 31 |
| | 10.7.1. Primary Endpoint | 31 |
| | 10.7.2. Secondary Endpoints | 33 |
| | CCI | |
| | 10.8. Pharmacokinetic Analysis | 41 |
| | 10.9. Safety Analysis | 41 |
| | 10.9.1. Adverse Events | 41 |
| | 10.9.2. Laboratory Variables | 42 |
| | 10.9.3. Vital Signs | 43 |
| | 10.9.4. Spirometry | 43 |
| | 10.9.5. Physical Examination | 43 |
| | 10.9.6. 12-Lead Electrocardiograms | 43 |
| 11. | CHANGES TO THE PROTOCOL SPECIFIED ANALYSIS DETAILED IN THE STATISTICAL A | ANALYSIS PLAN |
| 12. | REFERENCES | 45 |
| 13. | TABLES, FIGURES AND LISTINGS | 46 |
| | 13.1. Specific Presentation Details | 46 |
| | 13.2. List of Tables | 47 |
| | 13.3. List of Figures | 50 |

| ReV | iral Limited/REVD002 [hVIVO Services Ltd/VIR-CST-001] - CONFIDENTIAL 13.4. List of Listings | . 52 |
|---|---|---|
| 14. | TABLE AND LISTING SHELLS | |
| 15. | APPENDICES | 112 |
| | 15.1 Study VIR-CST-001 assay cut-offs and reporting | 112 |

# 1. STATISTICAL ANALYSIS PLAN APPROVAL FORM

| | | Signature | Date (ddmmmaaa) | Time<br>(hh:mm) | Local Time<br>Zone |
|---|---|---|---|---|---|
| | | | (ddmmmyyyy) | (nn:mm) | zone |
| Author(s): | | | | | |
| PPD | | | | | |
| Senior Statisticiar | l, | | | | |
| PPD | | | | | |
| Approval(s): | | | | | |
| PPD | | | | | |
| PPD | | | | | |
| ReViral, a Pfizer ( | ompany | | | | |
| | | | | _ | |
| PPD | | | | | |
| PPD | | | | | |
| hVIVO Ltd | | | | | |

# 2. STATISTICAL ANALYSIS PLAN AUTHOR



# 3. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|--------------|---------------------------------------------------|
| AE | Adverse event |
| ALP | Alkaline phosphatase |
| ALQ | Above the limit of quantification |
| ALT | Alanine transaminase |
| APTT | Activated partial thromboplastin time |
| AST | Aspartate transaminase |
| AUC | Area under the curve |
| BDR | Blind Data Review |
| BDRM | Blind Data Review Meeting |
| β-HCG | Beta human chorionic gonadotropin |
| BLQ | Below the level of quantification |
| BMI | Body mass index |
| BPM | Beats per minute |
| CI | Confidence interval |
| CK | Creatinine Kinase |
| Covid-19 | Coronavirus disease 2019 |
| CRF | Case Report Form |
| CRP | C-reactive protein |
| CSR | Clinical Study Report |
| DBP | Diastolic blood pressure |
| DP | Decimal places |
| ECG | Electrocardiogram |
| ET | Early termination |
| FEV1 | Forced expiratory volume in 1 second |
| FSH | Follicle-stimulating hormone |
| FU | Follow-up |
| FVC | Forced vital capacity |
| GGT | Gamma glutamyl transferase |
| GM | Geometric Mean |
| GSD | Geometric Standard Deviation |
| HbA1C | Glycated haemoglobin |
| HIV | Human immunodeficiency virus |
| HR | Heart Rate |
| HVC | Human Viral Challenge |
| hVIVO | hVIVO Services Limited |
| ICF | Informed consent form |
| IMP | Investigational medicinal product |
| INR | International normalised ratio |
| IQR | Inter-quartile range |
| ITT | Intention-to-Treat |
| ITT-I | Intention-to-Treat Infected |
| ITT-A | Intention-to-Treat Infected Analysis Population A |
| ITT-B | Intention-to-Treat Infected Analysis Population B |
| LDH | Lactate dehydrogenase |
| LRT | Lower respiratory tract |

| Abbreviation | Definition |
|--------------|--------------------------------------------------------------|
| MCH | Mean corpuscular haemoglobin |
| MCHC | Mean corpuscular haemoglobin concentration |
| MCV | Mean corpuscular volume |
| MedDRA | Medical dictionary for regulatory activities |
| NCI | New-onset chronic illness |
| PCR | Polymerase chain reaction |
| PD | Protocol deviation |
| PE | Physical examination |
| PEF | Peak expiratory flow |
| PFU | Plaque forming units |
| PK | Pharmacokinetic |
| PP | Per protocol |
| PT | Preferred term |
| PT | Prothrombin time |
| PTT | Partial thromboplastin time |
| RR | Respiratory rate |
| Q1 | Lower quartile |
| Q3 | Upper quartile |
| qicPCR | Qualitative integrative cycler polymerase chain reaction |
| qRT-PCR | Quantitative reverse transcription polymerase chain reaction |
| RBC | Red blood cells |
| RNA | Ribonucleic acid |
| RSV | Respiratory Syncytial Virus |
| SAE | Serious adverse event |
| SAP | Statistical analysis plan |
| SARS-CoV-2 | Sever acute respiratory syndrome coronavirus 2 |
| SBP | Systolic blood pressure |
| SD | Standard deviation |
| SE | Standard error |
| SOC | System organ class |
| SoE | Schedule of Events |
| SpO2 | Peripheral arterial oxygen saturation |
| TEAE | Treatment emergent adverse event |
| TFL | Tables, Figures and Listings |
| TSS | Total clinical symptoms |
| ULN | Upper limit of normal |
| ULOQ | Upper limit of quantification |
| URT | Upper respiratory tract |
| VL | Viral load |
| WBC | White blood cells |
| WHO | World Health Organisation |

# 4. INTRODUCTION

This statistical analysis plan (SAP) explains in detail the statistical analyses that will performed for the ReViral Limited study REVD002 [hVIVO study no: VIR-CST-001]. The analysis is outlined within the study protocol V3.0 (dated 31 October 2022) and this SAP contains a more technical and detailed description of those analyses. In particular, the SAP provides information on the definitions of the participant populations, analysis methods, and details the list of Tables, Figures and Listings (TFL) that will be produced by S-cubed Biometrics for use and inclusion within the Clinical Study Report (CSR). The SAP has been written and finalised before any unblinding of the study and prior to the database being locked.

Any deviations from the protocol specified analyses, and deviations from analyses stated within this SAP will be described within the CSR.

# 5. STUDY OBJECTIVES

# 5.1. Primary Objective

The primary objective is to assess the antiviral activity of RV299 compared to placebo in healthy adult participants infected with RSV-A Memphis 37b.

# 5.2. Secondary Objectives

- To evaluate the effect of RV299 compared to placebo in healthy adult participants inoculated with RSV in terms of antiviral effect assessed by:
  - o viral-load related endpoints;
  - o clinical symptom-related endpoints (using the 10 predefined symptoms in the graded symptom scoring system).
- To evaluate the effect of RV299 on nasal discharge in healthy adult participants inoculated with RSV when compared to placebo.
- To evaluate the safety of multiple orally administered doses of RV299 when compared to placebo.
- To monitor the safety of the challenge virus.
- To characterise the PK profile of RV299 after a single oral dose and after multiple oral doses in plasma from healthy participants inoculated with RSV.



### 6. STUDY DESIGN

## 6.1. Summary of Study Design

This is a single-centre, randomised, double-blind, placebo-controlled, proof-of-concept study in healthy adult male and female participants from 18 to 55 years of age, inclusive. The primary goal of this Phase 1b study is to assess the antiviral activity of RV299 against RSV in the viral challenge model. In addition, the safety, tolerability, and PK of RV299 will be assessed.

A total of 80 participants is planned to be enrolled in this study: 40 participants on RV299 and 40 participants on placebo.

The study is divided into the following study phases:

- Screening phase: from Day -90 to Day-3 pre-human viral challenge (HVC). Historical generic screening data collected through the hVIVO generic screening process may be transferred to this study after the study-specific consent form has been signed by the participant.
- Inpatient phase: Participants will be resident in the quarantine unit for approximately 15 days (from Day -2 to Day 12). Procedures will include:
  - o Pre-HVC:
    - Admission to guarantine unit on Day -2/-1.
    - Baseline assessments will be conducted as per Schedule of Events (SoE) up to Day
       0, pre-challenge.
  - HVC: RSV-A Memphis 37b virus inoculation on Day 0.
  - Post-HVC:
    - Randomisation to receive RV299 or matched placebo.
    - Administration of IMP (RV299/placebo). Each participant will receive IMP twice daily (~12 hours interval) for 5 consecutive days:
      - IMP dosing to start on confirmation of RSV infection, i.e., after a positive result by qualitative integrative cycler polymerase chain reaction (qicPCR). The qicPCR of nasal wash will be performed twice daily on Days 2-5 (Day 5 morning only), or until a positive result is received, whichever is sooner. The earliest start of IMP dosing will be in the evening of Day 2 post-HVC (IMP will be initiated 12 hours ± 1-hour post nasal wash confirmation of infection)

OR

- IMP would start in the evening of Day 5, if no positive result obtained by gicPCR
- Day 1 onwards and each day study assessments will be conducted as per SoE.
- Participants will be discharged from the quarantine unit on Day 12 (or may remain longer at the discretion of the principal investigator [PI]/investigator).
- Outpatient phase:
  - o Final visit: Day 28 (±3 days).

The overall study design is depicted in

| ReViral Limited/REVD002 [hVIVO Services Ltd/VIR-CST-001] - CONFIDENTIAL |
|-------------------------------------------------------------------------|
| Table 1. |

Table 1: Study Schematic: On-study Participant Progression

SCREENING INPATIENT PHASE: QUARANTINE/ISOLATION, HUMAN VIRAL OUTPATIENT PHASE

CHALLENGE, AND DOSING PHASE

| | - | | ī | | , | | - | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | Day 0 | | | | | |
| Day -90 to<br>Day -3<br>Screening* | | Day -2/-1<br>Admission<br>to<br>quarantine<br>unit | | Inoculation with challenge agent & assessments as per Schedule of Events | | Days 1 to 11 Dosing and assessments as per Schedule of Events | | Day 12<br>Discharge<br>from<br>quarantine<br>unit** | Follow-up<br>visit:<br>Day 28<br>(±3 days) |

### **NOTES:**

<sup>\*</sup>Screening assessments (including repeats, as required), may be performed up to Day -2/-1, defined as the first study day (quarantine admission) at the discretion of the PI/investigator and in accordance with the design of the study.

<sup>\*\*</sup>Release from quarantine is foreseen at Day 12 (12 days post inoculation) provided that, where appropriate, no virus is detected by qualitative virus antigen test or polymerase chain reaction (PCR) (negative virus antigen test or PCR below Ct cut-off) and the participant has no clinically significant symptoms. If the participant continues to have clinically significant symptoms and/or detectable virus on Day 12, additional extended quarantine stay may be required at the discretion of the Pl/investigator.

# 6.2. Randomisation / Treatment Allocation and Blinding

hVIVO assigns a unique 6-digit number to each participant in the hVIVO database. This number will be used to identify a participant up to the point of randomisation, on source documents, on all study correspondence, and in the study database. A separate randomisation number will be allocated to the participants at randomisation and will be used for allocation to a study arm. The randomisation number encodes the participant's assignment to 1 of 2 study arms (RV299/placebo) in a 1:1 ratio.

Randomisation numbers will be assigned sequentially in ascending order, and once assigned, that randomisation number will not be reassigned. The study site will keep a log of the randomisation number assigned to each participant.

A designated unblinded statistician, separate from the conduct or analysis of the study, will be responsible for the computer-generated randomisation schedule. Sealed copies of the randomisation code will be stored in a secure location.

Randomisation numbers will follow a 3-digit format e.g., 001. If participants are replaced as per Section 7.4, Participant Replacement Strategy, the replacement participant will be assigned a new, unique randomisation number equalling the randomisation number of the replaced participant, plus 100. This will ensure that the replacement participant receives the same allocated, blinded treatment as the participant who is being replaced.

A copy of the randomisation code list will be sent to the unblinded pharmacist/designee preparing the IMP, so that IMP can be prepared for each participant as appropriate. An independent statistician prepares the randomisation schedule, and the GMP pharmacy provider's pharmacy/designee will prepare the participant level IMP doses in line with the randomisation schedule.

Each participant will be dispensed blinded IMP, labelled with his/her unique randomisation number, throughout the study. With the exception of the unblinded pharmacist, unblinded IMP management personnel at the clinical site, the unblinded statistician preparing the randomisation code list, and the quality assurance auditors where necessary, the PI/investigator and all other clinical and nonclinical staff, (including the study statistician, data management staff), and the participants will remain blinded to the treatment allocation until after the database has been locked and approval for study unblinding has been given.

Following database lock, on receipt of authorisation from the Sponsor, a copy of the randomisation code list will be provided to the study statistician to conduct study unblinding for analysis.

#### 6.3. Time and Events Schedule

Details of the timing of study assessments and procedures can be found in Table 2.

Table 2: Schedule(s) of Events (SoE)

| Study Phase → | Screening<br>Phase* | | | | | (Quara | antine | Isolati | | ient Pha<br>Humar | | Challer | ıge [HV | 'C]) | | | | | Clinic Visit<br>Follow-up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day → | D -3 | | _ | | D 0 | | | | | | | | | | | 0 | | :<br>rge) | ys) |
| Procedure <b>♥</b> | D -90 to D | D -2 | 0-1 | Pre-HVC | FAC | Post-HVC | D 1 | D 2 | D 3 | D 4 | D 5 | 9 Q | D 7 | D 8 | 6 Q | D 10 | D 11 | D12<br>(Discharge) | D 28<br>(±3 days) |
| Vritten informed consent (a) | | | X | | | | | | | | | | | | | | | | |
| Eligibility criteria (+) | Х | | X | Х | | | | | | | | | | | | | | | |
| Medical & medication history | Х | | X | | | | | | | | | | | | | | | | |
| Demographics | Х | | | | | | | | | | | | | | | | | | |
| Height & body weight, body mass<br>ndex (BMI) (b) | Х | | X | | | | | | | | | | | | | | | (X) | (X) |
| Complete physical examination | Х | | X | | | | | | | | | | | | | | | Х | Х |
| Directed physical examination (incl. asal) | | | | (X) | | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | (X) | | |
| /ital signs (heart rate [HR], respiratory<br>ate [RR], systolic blood pressure [BP],<br>diastolic BP, oxygen saturation [SpO <sub>2</sub> ])<br>and tympanic membrane temperature | х | | Х | х | | | х | х | x | X | X | х | x | x | Х | х | х | Х | х |
| 12-lead ECG | Х | | X | | | | | | | | | | Х | | | | Х | | Х |
| Spirometry | Х | | | | | | | | | | | | | | | | | | |
| Patient Health Questionnaire (PHQ-9) | (X) | ( | X) | | | | | | | | | | | | | | | | |
| Generalised Anxiety Disorder<br>Questionnaire (GAD-7) | (X) | ( | X) | | | | | | | | | | | | | | | | |
| Alcohol breath test | X | | X | | | | | | | | | | | | | | | | Χ |
| Jrinalysis | Х | | X | | | | | | | | | | | | | | | Х | Х |
| Jrine drugs of abuse and cotinine screen | Х | | X | | | | | | | | | | | | | | | | Х |
| Jrine pregnancy test | Х | | | | | | | | | | | | | | | | | Х | Х |
| Symptom diary card (c) | | (X) | 3X | | 3X | | 3X | 3X | 3X | 3X | 3X | 3X | 3X | 3X | 3X | 3X | 3X | Х | |
| 24-hour paper tissue collection & nasal<br>discharge weight (d) | | | Х | х | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | |

| Study Phase → | Screening<br>Phase* | | | | | (Quara | antine | Isolatio | • | ient Ph<br>Humaı | | Challer | ıge [HV | ′C]) | | | | | Clinic Visit<br>Follow-up | wal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day → | D -3 | | DO DO COMPANDO DO | | | | | | | | | | | | s<br>ys) | Early Withdrawal | | | | |
| Procedure <b>♥</b> | D -90 to D | D-2 | 0-1 | Pre-HVC | HVC | Post-HVC | 10 | D 2 | D 3 | D 4 | D 5 | D 6 | D 7 | D 8 | 6 Q | D 10 | D 11 | D12<br>(Discharge) | D 28<br>(±3 days) | Early V |
| Product Administration | | | | | | | | <u>I</u> | | | I. | | | | | | | | | |
| Randomisation | | | | | | | | (X) | (X) | (X) | (X) | | | | | | | | | |
| RSV299/placebo dosing (k) | | | | | | | | (X) | (2X) | (2X) | (2X) | (2X) | (2X) | (2X) | (2X) | (X) | | | | |
| Challenge virus inoculation | | | | | Х | | | | | | | | | | | | | | | |
| Collection Of Blood Samples | | | | | | | | | | | | | | | | | | | | |
| Serum follicle-stimulating hormone (FSH) (post-menopausal women) | Х | | | | | | | | | | | | | | | | | | | |
| Serum β-human chorionic<br>gonadotrophin (β-hCG) pregnancy test<br>(all females) | | , | × | | | | | | | | | | | | | | | | | |
| Hepatitis B, & C, human immunodeficiency virus (HIV) serology | Х | | | | | | | | | | | | | | | | | | | |
| Blood Pharmacokinetics (e) | | | | | | | | (X) | (X) | (X) | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Haematology (f) | Х | ) | X | | | | | | | | | | Х | | | | Х | | Х | Х |
| Biochemistry (f) | Х | ) | X | | | | | | | | | | Х | | | | Х | | Х | Х |
| Coagulation | Х | | | | | | | | | | | | | | | | | | | |
| Cardiac enzymes | Х | ) | X | | | | | _ | | _ | | _ | Х | | _ | | Х | | | |
| Thyroid function test | Х | | | | | | | | | | | | | | | | | | | |
| CCI | | | | | | | | | | | | | | | | | | | | |
| | | ) | X | | | | | | | | | | | | | | | | | |

| Study Phase → | Screening<br>Phase* | | | | | (Quara | antine | Isolatio | - | ient Ph<br>Humaı | | Challen | ge [H\ | /C]) | | | | | Clinic Visit<br>Follow-up | wal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Day <b>→</b><br>Procedure <b>↓</b> | D -90 to D -3 | D-2 | D-1 | Pre-HVC | HVC D0 | Post-HVC | D 1 | D 2 | D 3 | D 4 | D 5 | D 6 | D 7 | D 8 | 6 0 | D 10 | D 11 | D12<br>(Discharge) | D 28<br>(±3 days) | Early Withdrawal |
| Collection Of Respiratory Samples | | | | | | | | | | | | | | | | • | | | | |
| Nasopharyngeal swab - respiratory pathogen screen incl. SARS-CoV-2 (h) | | ) | × | | | | | | | | | | | | | | | | | |
| Nasopharyngeal swab- RSV discharge test | | | | | | | | | | | | | | | | | (X) | (X) | | |
| CCI | | | I | | | | | | | | | | | | | | | | | |
| qicPCR (i) | | | | | | | | 2X | 2X | 2X | Х | | | | | | | | | |
| Safety Assessments | | | | | | | | | | | | | | | | | | | | |
| Adverse event (AE) recording (j) | | • | | | | | | | | | | | | | | | | | - | Х |
| Concomitant medications (j) | | 4 | | | | | | | | | | | | | | | | | - | Х |

# **KEY NOTES FOR TIME AND EVENTS SCHEDULE:**

| (X) | The assessment may be optional, or at the PI's discretion. The PI may perform additional safety assessments as required. |
|---|---|
| Х | Once daily, at approximately the same time each day, where applicable. |
| 2X | Twice daily (~12 hours between assessments [± 1 hour]). |
| 3X | Three times daily (at the same times each day [± 1 hour]). |
| * | Potential participants will be screened using the hVIVO generic screening process, and individuals who pass this screen will be admitted to the quarantine unit 1 to 2 days before challenge with study virus and provide study-specific informed consent. They will then be screened for eligibility for this study before viral challenge on Day 0. Results of tests or examinations performed under hVIVO generic screening process may be used to determine eligibility without the need to repeat the assessment if it is within 28 days prior to viral challenge/dosing with IMP. |
| + | Only the applicable inclusion/exclusion criteria will be reviewed at each time point. |
| а | Study-specific consent may occur on the day of admission, providing all required eligibility information has been collected through the Health Research Authority -approved hVIVO generic screening process. |

| b | Height will be taken at screening only. |
|---|---|
| С | After the baseline has been set, assessments will be performed at the same time each day (±1 hour from baseline) during quarantine. • Symptom diary card baseline: Day -1 (measurements on this day will be taken approximately 8 hours apart, ±1 hour). • Nasal wash baseline: Day 2 (sampling will be performed approximately 12 hours apart, ±1 hour). |
| d | Distribution of paper tissues and bags will start on Day -1, with the first collection on Day 0. Thereafter, collection of paper tissues will occur at the same time each day (±1 hour) with tissues distributed 24 hours ahead. |
| е | <ul> <li>Blood Pharmacokinetics: plasma samples for RV299 assay will be collected as follows:</li> <li>First dose (Dose 1): 0.5 hours pre-dose, and at the following hours post-first dose: 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84 and 96 hours (note samples taken up to and including 10 hours post-dose should be taken at the indicated time point ±5 minutes. Samples taken thereafter at 12, 24, 36, 48, 60, 72, 84, and 96 hours post-first dose should be taken within the 30 minutes before the next IMP intake).</li> <li>Last dose (Dose 10): 0.5 hours pre-dose, and at the following hours post-last dose: 1, 1.5, 2, 2.5, 3, 4, 5, 6, 7, 8,10, 12, 24, 36, 48, 60, 72, 84, and 96 hours (note samples taken up to and including 10 hours post-dose should be taken at the indicated time point ±5 minutes; samples taken thereafter should be taken at the indicated time point ±30 minutes).</li> <li>For participants who started dosing on Day 4, am, onwards, the 60-hour, 72-hour, 84-hour, or 96-hour timepoints after Dose 10 could occur after the participant has met the discharge criteria on Day 12. Thus, for a subset of participants, these timepoints could be after discharge. The guidance for the 60-hour, 72-hour, 84-hour, and 96-hour PK sample collection is as follows:</li> <li>For participants who started dosing on Day 4, am, onwards, and who meet the discharge criteria on Day 12, the 60-hour, 72-hour, 84-hour, and 96-hour timepoint samples may be omitted, as applicable, if it occurs after discharge.</li> <li>For participants who started dosing on Day 4, am, onwards, and who do not meet the discharge criteria on Day 12 the 60-hour, 72-hour, 84-hour, and 96-hour PK timepoint samples should be collected up to the point where participant meets the discharge criteria.</li> </ul> |
| f | Blood will be drawn under non-fasted conditions. Repeat bloods may be drawn under fasted conditions if a lipid profile (triglyceride) or glucose is required (at the PI's discretion). All participants will be dosed under fasted conditions. For all doses, a pre-dose and post-dose fasting period of 0.5 hour to 1 hour applies. No fluid intake (including water) is allowed for 1 hour pre-dose to 1-hour post-dose). |
| g | Virus serology (RSV neutralisation antibody assay) will be performed to determine eligibility and seroconversion. |
| h | Upper respiratory tract swab (e.g., nasopharyngeal swab, mid-turbinate swab, oropharyngeal swab) for respiratory virus screen to assess for the presence of respiratory pathogen if found positive for any pathogen in the panel, the participant will not be eligible for the current quarantine. |
| i | Post inoculation nasal wash virology samples will be collected at the same time each day during quarantine (± 1 hour from baseline on Day 2) and used for qRT-PCR and viral culture assay (as appropriate). Samples may be used for related viral genomics samples collected between the morning of Day 2 and the morning of Day 5 will also be used for qicPCR until a positive result is received (to support triggered dosing). |
| j | Adverse events and concomitant medications are reviewed throughout the study including pre- and post-dosing with IMP and pre- and post-RSV virus inoculation. |

# ReViral Limited/REVD002 [hVIVO Services Ltd/VIR-CST-001] - CONFIDENTIAL

| k | IMP doses as oral solution/suspension will be taken with 140 mL of water (50 mL water rinse of IMP bottle following administration, and 90 mL post-dose). |
|---|---|
| | All participants will be dosed orally, in the seated position, under fasted conditions, under the direct supervision of the investigator (or delegate), and in accordance with the randomisation schedule. Each participant will receive IMP twice daily (~12 hours interval) for 5 consecutive days, in total 10 doses, IMP dosing to start on confirmation of RSV infection. The earliest start of IMP dosing will be in the evening of Day 2 post-HVC or IMP dosing will start in the evening of Day 5, if no confirmation of RSV infection. |
| Note: | Parenthesis indicates the assessment may be optional, or at the PI's discretion. |
| | The PI/investigator may perform additional safety assessments as required. |
| | Where any nasal sampling time points occur together, the order of sampling will typically be (1) nasopharyngeal swab followed by (2) nasal wash. |

Statistical Analysis Plan Page 19 of 113 Version 01-00, 20DEC2022

# 6.4. Interim Analysis / Data Monitoring

No interim analysis (i.e., an analysis of early trial data, before enrolment is completed, to detect trends that might warrant modification of the protocol, change in data being collected or trial termination) is planned for the study.

### 7. STUDY ENDPOINTS

# 7.1. Primary Endpoint

The primary endpoint is:

The area under the curve (AUC) for RSV viral load measured in nasal washes by quantitative real time reverse transcription polymerase chain reaction (qRT-PCR) in participants inoculated with RSV-A Memphis 37b, starting at initial administration of investigational medicinal product (IMP) up to planned discharge from quarantine (Day 12, am).

## 7.2. Secondary Endpoints

The secondary endpoints are:

- Additional viral load endpoints relating to antiviral effect include but are not limited to:
  - Peak viral load of RSV as defined by the maximum viral load determined by qRT-PCR measurements in nasal samples starting from initial administration of IMP up to planned discharge from quarantine (Day 12, am).
  - Time (days) to confirmed negative test by qRT-PCR measurements in nasal samples starting at initial administration of IMP to first confirmed undetectable assessment after peak measure.
  - Time (days) to confirmed negative test by qRT-PCR measurements in nasal samples starting from peak qRT-PCR after initial administration of IMP to first confirmed undetectable assessment after peak measure.
  - Time (days) to peak qRT-PCR in nasal samples, starting from initial administration of IMP.
  - Area under the viral load-time curve (VL-AUC) of RSV challenge virus as determined by viral culture on nasal samples, starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am).
  - Peak viral load of RSV as defined by the maximum viral load determined by viral culture measurements in nasal samples starting from initial administration of IMP up to planned discharge from quarantine (Day 12, am).
  - Time (days) to confirmed negative test by viral culture measurements in nasal samples starting at initial administration of IMP to first confirmed undetectable assessment after peak measure.
  - Time (days) to confirmed negative test by viral culture measurements in nasal samples starting from peak viral culture after initial administration of IMP to first confirmed undetectable assessment after peak measure.
  - Time (days) to peak viral culture in nasal samples, starting from initial administration of IMP.
- Clinical symptom-related endpoints include, but are not limited to:
  - Area under the curve over time of total clinical symptoms (TSS-AUC) as measured from 10 symptoms within the graded symptom scoring system collected 3 times daily starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am).
  - Area under the curve over time of total clinical symptoms change from baseline (TSS-AUCCFB) as measured from 10 symptoms within the graded symptom scoring system

- collected 3 times daily starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am).
- Peak symptoms diary card score: peak total clinical symptoms (TSS) as measured from 10 symptoms within the graded symptom scoring system collected 3 times daily starting from initial administration of IMP up to planned discharge from quarantine (Day 12, am).
- Peak daily symptom score: individual maximum daily sum of symptom score from initial administration of IMP up to planned discharge from quarantine (Day 12, am).
- Time (days) to symptom resolution as measured from 10 symptoms within the graded daily symptom scoring system starting at initial administration of IMP to time of returning to baseline score.
- Time (days) to symptom resolution as measured from 10 symptoms within the graded daily symptom scoring system starting at peak symptoms after initial administration of IMP to time of returning to baseline score.
- Time (days) to peak as measured from 10 symptoms within the graded daily symptom scoring system starting from initial administration of IMP to the time of peak daily symptom score.
- Total weight of mucus produced starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am).
- Total number of tissues used by participants starting at initial administration of IMP up to planned discharge from quarantine (Day 12, am).
- Safety data including, but not limited to:
  - Occurrence of adverse events (AEs) from initial administration of IMP up to the Day 28 follow-up.
  - Occurrence of serious AEs (SAEs) from initial administration of IMP up to the Day 28 followup.
  - Occurrence of AEs related to the viral challenge from viral challenge (Day 0) up to the Day 28 follow-up.
  - Occurrence of SAEs related to the viral challenge from viral challenge (Day 0) up to the Day 28 follow-up.
  - Use of concomitant medications from viral challenge (Day 0) up to the Day 28 follow-up.
- Secondary endpoints related to PK include, but are not limited to:
  - Time to maximum plasma concentration  $(t_{max})$ , terminal half-life  $(t_{1/2})$ , maximum observed plasma concentration  $(C_{max})$ , area under the plasma concentration-time curve from time zero to the end of the dosing interval  $(AUC_{\tau})$ , area under the plasma concentration-time curve over the last 24 hours dosing interval  $(AUC_{0-24h})$  and area under the plasma concentration-time curve from time zero to infinity  $(AUC_{0-\infty})$ .



CONFIDENTIAL

hVIVO Services Ltd/VIR-CST-001

| CCI | | | |
|-----|------|---|------|
| | <br> | | <br> |
| | | 1 | |

### 9. STUDY POPULATIONS

Populations defined below will be reviewed against the study database at a blinded data review meeting (BDRM). The database at this time will be nearly final (i.e., the meeting may result in further data queries/changes post meeting), so inclusion/exclusion of participants from populations defined at this meeting will be further checked (post meeting) against a final locked database and will then be finalised prior to unblinding.

## 9.1. Intent-to-Treat (ITT) Population

The intent-to-treat (ITT) population will consist of all randomised participants who received challenge virus and at least 1 dose of IMP. Participants will be analysed in the treatment group they were randomised to.

## 9.2. Intent-to-Treat Infected (ITT-I) Population

The intent-to-treat infected (ITT-I) population will consist of all randomised participants who received challenge virus and at least 1 dose of IMP, and meet the criterion for RSV infection. Participants will be analysed in the treatment group they were randomised to.

As per Section 10.7.2 in the protocol, a laboratory-confirmed RSV infection requires one or both of the following definitions to be met:

- At least 2 positive detections by viral load qRT-PCR assay specific for the challenge virus, reported on 2 consecutive days;
- One positive detection by viral load qRT-PCR assay, specific for the challenge virus, in which an
  aliquot of the same sample has also tested positive in a viral culture assay appropriate for
  detecting the challenge virus.

For qRT-PCR and the viral culture assay a positive detection is any positive numeric or "detected" value.

# 9.3. Intent-to-Treat Infected Analysis Population A (ITT-A) Population

The intent-to-treat infected analysis population A (ITT-A) population will consist of all randomised participants who received challenge virus and at least 1 dose of IMP, and meet the criterion for laboratory-confirmed RSV infection as defined for the ITT-I, using only assessments <u>prior to</u> taking IMP. Participants will be analysed in the treatment group they were randomised to.

The assessments prior to taking IMP includes all qRT-PCR assessments performed before dosing, including the assessment immediately before dosing. In addition, if the infection was seen (via a positive qRT-PCR value) before dosing but the confirmatory value (as per the first part of the viral shedding definition in Section 10.7.2 of the protocol) was taken after dosing, then the participant will be declared as infected before IMP administration, and hence will form part of the ITT-A Population.

Note: The assessments prior to dosing with IMP will include all qRT-PCR and viral culture assessments performed on samples collected before dosing, including the sample collected immediately prior to dosing.

# 9.4. Intent-to-Treat Infected Analysis Population B (ITT-B) Population

The intent-to-treat infected analysis population B (ITT-B) population will consist of all randomised participants not already in the ITT-A Population, who received challenge virus and at least 1 dose of IMP, and meet the criterion for laboratory-confirmed RSV infection as defined for the ITT-I, using only assessments <u>after</u> taking IMP. Participants will be analysed in the treatment group they were randomised to.

Note: The assessments after dosing with IMP will include all qRT-PCR and viral culture assessments on samples that are collected after dosing and will not include the sample collected immediately prior to dosing.

# 9.5. Per Protocol (PP) Population

The per-protocol (PP) population will consist of all ITT-I population participants who have no major protocol deviations, and who completed the quarantine period up to the final day of quarantine (Day 12) and received all 10 doses of IMP. Participants will be analysed in the treatment group they were randomised to.

# 9.6. Safety Population

The safety population will consist of all randomised participants who received challenge virus and at least 1 dose of IMP. Participants will be analysed according to the treatment they received.

# 9.7. PK Population

The PK population will consist of all ITT population participants with at least one post-dose PK result. Participants will be analysed according to the treatment they received.

## 10. PLANNED STATISTICAL METHODS

#### **10.1.** Statistical Considerations

#### 10.1.1. General Definitions

In all applicable summary/analysis presentations of safety endpoints, Baseline is defined as the last non-missing assessment value for a participant, for that particular parameter, that is prior to inoculation of challenge virus, unless over-ruled after review of data at the BDRM or otherwise stated in the appropriate endpoint sections below, whatever the reason for that assessment (e.g. if it is a repeat assessment, then it should be used as the baseline). For efficacy endpoints, the baseline definition is as per the appropriate endpoint sections below. For the derivation of most efficacy endpoints, the first assessment to be used should be the assessment that was taken at the time of first administration of IMP. For example, if a participant was first dosed on the morning of Day 3 then the first qRT-PCR value to be used in the AUC of qRT-PCR viral load (from time of first administration) derivation should be the Day 3 morning assessment. For endpoints using symptom diary card data, the definition of baseline will be defined in greater detail within the appropriate sections of the SAP.

A participant will be classed as infected, and therefore randomised to be dosed, when they have a positive result for RSV-A Memphis 37b by qualitative integrative cycler polymerase chain reaction (qicPCR) from nasal wash sample. IMP administration will be initiated 12 hours after a positive result. However, if a participant remains uninfected, IMP administration will begin on the evening of Day 5.

For participants that extend their time in quarantine beyond Day 12, the additional assessments beyond Day 12 will be listed only, and will not be used for the derivation of any efficacy endpoints. For the avoidance of doubt, the assessment performed on the morning of Day 12 will be the final assessment used for all analyses and summaries for all participants. If additional assessments are taken on Day 12, then they will be listed only. However, the use of data beyond the morning of Day 12 will be discussed at the BDRM.

A participant will be considered to have completed the study after their attendance at the last planned study visit (Day 28 (+ 3 days)), or the last unscheduled visit (if any occur), as applicable.

Data recorded for replaced participants will be listed. However, these participants will only be included in tables where they meets the inclusion criteria for the relevant population.

Within summary presentations/analyses it is envisaged that only scheduled protocol visit values will be used for post-baseline time points and unscheduled visits will not be summarised in tables. All unscheduled visits will be listed. However, at the BDRM the occurrence of such non-scheduled data will be reviewed for each participant to decide if (and how) any such data point(s) should be included within summary presentations/analyses. Any such decisions will be documented in the BDRM minutes.

For assessments made on Day 0 (either pre or post challenge), the date and time of inoculation will be compared to the date and time of assessment to ensure they are assigned to either pre or post challenge accurately.

### 10.1.2. Data Presentation

The specific format and content of each data presentation is shown in Section 

Summary tables will be presented by treatment group. For demographic, baseline, and safety data these will also be summarised for all participants.

Within all Tables and Figures, the treatment groups will be labelled and ordered as follows:

- RV299
- Placebo
- Overall (including RV299 and placebo participants, for demographic, baseline and safety data)

The scheduled protocol visits will be labelled in report presentations as follows:

- "Admission (Day-2/Day-1)"
- "Day 0 (pre-HVC)"
- "Day 0 (HVC)"
- "Day 0 (post-HVC)"
- "Day x" (where x=1 to 12)
- "Follow-up (Day 28)"
- "Early Withdrawal"

As the study day of IMP administration day will differ between participants, "x Days from IMP Administration" (where x=0 to 11) will be presented for efficacy outputs relating to clinical symptoms and PK. These assessments should be presented in relation to the IMP administration, rather than the inoculation day.

For data with multiple assessments on one study day, each assessment will be numbered sequentially (e.g. Assessment 1, Assessment 2 etc.) and will be relative to the first administration of IMP. Further details will be provided in the relevant sections of the SAP.

Within some tables, only "Baseline" may be shown (as applicable) instead of the scheduled visits Day 0 (pre-HVC) and Day-2/Day-1 (with baseline being chosen as defined in Section 10.1.1 and in the relevant endpoint sections).

Where duplicate information is collected on both the database and on the vendor data transfer(s) (e.g., sampling date and time) this information will be reconciled by data management and then the information from the vendor data transfer(s) will be included in Participant Listings.

All variables will be listed to the same number of decimal places as reported. Continuous endpoints will be summarised by: n, n missing, mean, standard deviation (SD), %CV, median, lower quartile (Q1), upper quartile (Q3), minimum (Min) and maximum (Max). Where appropriate, 95% confidence intervals (CIs) for the mean and/or median may be presented. For selected summaries the geometric mean (GM) and geometric standard deviation (GSD) will also be presented to aid interpretation. The SD will only be presented in summaries where the corresponding n is greater than or equal to 3.

The number of decimal places (DP) each summary statistic is rounded to for display in the summary tables, relative to the number of DP the parameter is recorded to, is shown in Table 3.

Table 3: Number of decimal places to use to display each summary statistic.

| Statistics | Number of DP for display |
|--------------------------|--------------------------|
| Min, Max | Same as recorded |
| Mean, GM, Median, Q1, Q3 | 1 more DP than recorded |

SD, GSD, %CV, 95% CI

2 more DP than recorded

For endpoints that require a geometric mean to be produced, and those endpoints can have raw values of 0 (zero), the GM calculation will add an appropriate constant value to all raw values prior to logging and will subtract that constant value from the final calculated anti-logged mean. The constant value used will be documented in the footnote of the tables. The value is typically 1 however it may be another small value which is in line with the scale of the data should a value of 1 be unsuitable. The GM and GSD are calculated as follows:

```
GM = anti-log ( mean ( log_{10} ( endpoint values + constant ) ) ) - constant GSD = anti-log ( SD ( log_{10} ( endpoint values ) ) )
```

The %CV will be calculated as %CV = 100 \* (SD / mean) using untransformed values.

Categorical variables will be summarised using proportions (counts and percentages). The specific approach to calculating percentages (relevant denominator) is detailed within each (relevant) Table template (Section ).

All collected data will be included within participant listings.

# 10.1.3. Early Withdrawal Visit

If a participant withdraws prior to Day 28 they will complete an early withdrawal visit. The data collected at this visit will be summarised as the nearest scheduled visit, unless the nearest visit already has data, in which case it will be summarised as the next scheduled visit. The data collected at the early withdrawal visit will be listed as the early withdrawal visit.

For example, if a participant withdraws at the Day 8 visit the data collected at the early withdrawal visit will be included in the summaries of Day 8. If, however, the participant withdrew between Day 8 and Day 9, after attending as normal on Day 8, the data collected at their early withdrawal visit will be included in the Day 9 summaries.

# 10.1.4. Statistical Testing and Estimation

Statistical analyses for the primary and secondary endpoints will be performed using appropriate two-sided hypothesis tests at the 5% significance level.

For continuous data, an analysis of covariance (ANCOVA) will be used to compare means between the RV299 and placebo groups. The ANCOVA will have treatment group as a fixed effect and baseline viral load as a covariate, unless stated otherwise in the relevant endpoint section. Should data not satisfy the assumptions, an appropriate alternative test, e.g., Wilcoxon Rank-Sum test will be used.

P-values will be rounded to 4 decimal places. All p-values that round to 0.0000 will be presented as <0.0001 and p-values that round to 1.000 will be presented as >0.9999.

# 10.1.5. Handling of Dropouts or Missing Data

No imputation methods will be used to manage the occurrence of missing data. Only observed data at each scheduled visit will be reported.

For adverse events and concomitant medications the approach to handle missing data has been described in Sections 10.9.1 and 10.5 respectively. For any other data which has partial dates, these dates will be completed using a suitably conservative approach.

Any other mechanisms to adjust for missing data will be outlined within the relevant endpoints section.

## 10.1.6. Interim Analysis and Data Monitoring

No interim analyses are planned to be performed.

## 10.1.7. Multiple Comparison/Multiplicity

As this is an early phase study, no adjustments will be made to address multiplicity.

# 10.1.8. Model Checking and Sensitivity Analyses

Statistical hypothesis testing will be presented using parametric tests where an ANCOVA will be the preferred statistical method. However, if the parametric test assumptions fail, non-parametric alternatives will be presented.

The normality of the error term from fitted models will be checked by performing the Shapiro-Wilk's test of normality of the residuals and producing normality probability plots of the residuals.

For cases where the normality assumption fails to hold, the treatment effect will be assessed by the non-parametric Wilcoxon rank-sum test.

# 10.1.9. Data Conversion (CDISC)

For the reporting of this study there is no requirement for CDISC SDTM and/or ADaM standards to be applied.

# 10.1.10. Software

Data will be reported using SAS version 9.4 (SAS Institute Inc, Cary, North Carolina, USA).

## 10.2. Participant Disposition

The number of participants enrolled (signed ICF), the numbered receiving challenge agent inoculation, the number randomised, the number receiving at least one dose of IMP and receiving all doses of IMP, the number discontinuing IMP early, the number withdrawing from the study, those completing the study (Day 28 visit), and the numbers in each population will be summarised for all participants and by treatment group. The reasons for early discontinuation of IMP and reasons for withdrawal from the study will also be summarised by treatment group.

A listing will be provided including details of informed consent, randomisation and quarantine admission.

#### 10.3. Protocol Deviations

Participants data will be reviewed for major protocol deviations by a qualified clinical reviewer prior to database lock and unblinding, at the BDRM. Participants with any major protocol deviations will be documented within the BDRM minutes, and such participants will be excluded from the PP population.

All protocol deviations will be listed.

# 10.4. Demographic and Other Baseline Characteristics

The safety population will be used in summaries of demographic and baseline data. No statistical testing will be used to compare treatment groups for different baseline characteristics.

## 10.4.1. Demographics

Demographic variables collected at Screening; sex, age, ethnicity, race, height (cm), weight (kg) and body mass index (BMI) will be summarised by treatment group and across all participants.

Age at screening and BMI are recorded in the database and do not need require derivation.

## 10.4.2. Substance Use History and Recreational Drugs of Misuse

Substance use history and any recreational drug misuse will be collected at screening and listed for all participants.

## 10.4.3. Reproductive Status and Contraceptive Use

The reproductive status and use of contraception will be collected at screening and listed for all participants.

## 10.4.4. Medical History

Medical history data will be coded using MedDRA, Version 25.0 (March 2022) and all data will be listed.

#### 10.5. Prior and Concomitant Medications

Prior and concomitant medication terms will be coded using the World Health Organisation (WHO) Drug Dictionary Enhanced (WHO Drug Global, Version March 1 2022). A medication will be assigned as being prior to inoculation based on the start and stop dates of the medication and the date of challenge agent inoculation. If the medication stop date is before the inoculation date, the medication will be assigned as being prior to inoculation. A medication will be assigned as being prior to IMP or concomitant with IMP, based on the start and stop dates of the medication and the IMP. If the medication stop date is before the IMP start date and after the date of inoculation, the medication will be assigned as being prior to IMP. In all other situations, the medication will be assigned as being concomitant with IMP. If a participant has separate periods of taking specific medications, then that medication is only counted once within the specific period of observation (i.e., prior, or concomitant) where it is taken.

Note: Start and Stop times will not be used for determining if a medication is concomitant or not.

Concomitant medications up to the Day 28 visit will be summarised, using the Safety Population, by treatment group (and across all participants), Drug Class (L3) and preferred base name (01001). If Level 3 is missing for a medication then Level 2 will be used instead.

Prior medications will not be summarised but these will be listed.

## 10.6. IMP Exposure and Compliance

The study consists of 10 doses of IMP administered twice daily for 5 consecutive days. The expected number of doses will be calculated using the start/stop dates and times for each participant. Compliance with IMP will be derived as:

(number of doses received/number of doses expected) \* 100.

Compliance will be summarised by treatment group and for all participants as a continuous variable and will also be summarised categorically in the following classifications: <80%, 80-120% and >120%.

### 10.7. Statistical Analysis

All efficacy analyses will be based on the ITT-I population as the primary analysis. Where the populations differ to ITT-I population by 1 participant within a treatment group, the primary and selected secondary analyses will be repeated for the ITT-A, ITT-B, ITT and PP populations. This will be reviewed and documented at the BDRM.

# 10.7.1. Primary Endpoint

# 10.7.1.1 Main Analysis

The primary endpoint is the AUC of RSV-A Memphis 37b viral load measured in nasal washes by qRT-PCR, from the last measurement collected prior to the first administration of IMP until the last measurement collected up to the morning of Day 12 (Quarantine discharge). The viral load data will be supplied as log<sub>10</sub> copies/mL and will be used for this main analysis and to calculate the AUC using the trapezoidal rule [1].

The AUC will be summarised for RV299 and placebo using descriptive statistics and an ANCOVA with treatment group as a main effect and the baseline value as a covariate. The baseline value will be the qRT-PCR viral load value from the last measurement collected prior to the first administration of IMP. The treatment comparison will be presented, including the LS mean treatment difference with the corresponding two-sided 95% confidence interval and p-value. The equivalent Wilcoxon rank-sum tests will be provided in place of the ANCOVA where the assumptions of the parametric test are not met.

As nasal washes are scheduled to be taken twice daily for Days 2 to 11 (and once on Day 12), in order to calculate the AUC, the actual time that the assessment was collected will be used within the AUC calculation. The AUC calculation will be based on the available non-missing assessment values between the start and end of the defined AUC time period. However, for an AUC to be derived, a participant should have at least one non-missing data recording at the start of the AUC period (e.g. date of first administration of IMP) and also at the end of the AUC time period (e.g. Day 12). In addition, the participant should have at least 1 non-missing data recording on each day between the start and end of the defined AUC time period (i.e. at least 1 out of the 2 possible assessments on each Day)). Any missing data will be reviewed at the BDRM, for its potential impact on this endpoint, and any decisions to exclude participants as a result of these criteria will be documented in the BDRM minutes. For the reporting of AUC, where appropriate, qRT-PCR values that are 'Not Detected' or 'Detected' will be reassigned using the substitution values shown in the table in Appendix 15.1.

As well as a descriptive statistics summary of AUC values, the mean qRT-PCR values (+/- 1 Standard Error (SE)) will be displayed graphically by day (relative to first dose of IMP) and assessment, and treatment group. In order to calculate the time point that each assessment will be presented against,

a relative day and relative assessment will be assigned. The last qRT-PCR measurement collected prior to the first dose of IMP will be assigned to be the value at time point 1, while measurements collected on subsequent assessments and days will be assigned to subsequent time points in sequential order (i.e. time point 2, 3 and so on). Time point 1 will be presented against Day 0 assessment 1, while subsequent time points will be presented against Day 0 assessment 1, and so on.

[Line graph: y-axis = mean of qRT-PCR ( $log_{10}$  copies/mL), x-axis = day relative to dosing, one line for each treatment on same plot].

A boxplot will also be presented by day (relative to first dose of IMP) and assessment, plotting the median and mean qRT-PCT values for each treatment group, with the corresponding summary statistics.

[Box plot: y-axis = mean of qRT-PCR ( $log_{10}$  copies/mL), x-axis = day relative to dosing, one box-and-whisker for each day, with each treatment panelled with RV299 at the top and placebo below].

Note: For multiple assessments taken within each day, so as to be able to plot mean values across participants (within a treatment group) by day, the actual collection time point (which may differ across participants) will not be used. Rather all first and second assessments will have mean values separately calculated and plotted as two means within each day. These two means will be shown equally spaced along the x-axis within the graph.

## 10.7.1.2 Sensitivity Analyses

- 1. The first sensitivity analysis of the AUC of RSV viral load measured in nasal washes by qRT-PCR will be presented for a fixed time period, from the last measurement collected prior to the first administration of IMP to the scheduled assessment occurring 6.5 days afterwards (e.g. if a participant does not have a positive qicPCR then they will be dosed on Day 5 (evening) and they will be followed up to the morning of Day 12 with 14 assessments in total) which represents the AUC over the longest possible time period over which all subjects are sampled.
- 2. A second sensitivity analysis of the AUC of RSV viral load measured in nasal washes by qRT-PCR will be presented for a fixed time period, which will include data from the morning assessment on Day 2 (i.e. the first qRT-PCR assessment measured) through to the morning of Day 12.
- 3. A third sensitivity analysis of the AUC of RSV viral load measured in nasal washes by qRT-PCR, from the last measurement collected prior to the first administration of IMP until the last measurement collected up to the morning of Day 12 (Quarantine discharge), will be presented where the AUC will be calculated using unlogged viral load data (i.e. the supplied value will be anti-logged to get a value as copies/mL).

The AUC analyses will be summarised by treatment group. The same statistical testing methods as applied to the main analysis of the primary endpoint will be applied to each sensitivity analysis. For the third sensitivity analysis, the data will be log-transformed (base 10) prior to statistical analysis.

## 10.7.2. Secondary Endpoints

# 10.7.2.3 Viral Load Endpoints

Peak Viral Load of RSV as Defined by the Maximum Viral Load Determined by qRT-PCR Measurements in Nasal Samples Starting from Initial Administration of IMP up to Planned Discharge from Quarantine

Using the scheduled protocol assessments from the last measurement collected prior to the first dose of IMP to morning of Day 12 (Quarantine discharge), the highest qRT-PCR viral load value observed in nasal samples for each participant will be summarised and analysed in a similar fashion to the primary efficacy endpoint described in Section 10.7.1.

Participants who stay undetectable (i.e. a 'Not Detected' value) during quarantine will be replaced with the 'Not Detected' value shown in the table in Appendix 15.1.

Time to Confirmed Negative Test by qRT-PCR Measurements in Nasal Samples Starting from Initial Administration of IMP to First Confirmed Undetectable Assessment after Peak Measure

The time from the first administration of IMP to the first confirmed negative qRT-PCR test after the peak qRT-PCR measurement will be calculated in days as:

Date and time of first confirmed negative test after peak qRT-PCR measurement – Date of and time of first IMP administration.

A negative test is defined as two consecutive 'Not Detected' results in the qRT-PCR test, with the date and time of the first negative test being utilised in the calculations. The peak qRT-PCR is defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who did not have a confirmed undetectable assessment after first administration of IMP are censored at their last detectable assessment after their peak qRT-PCR measurement. Participants who stay undetectable during quarantine will be excluded from this analysis. Participants who return a positive result after two consecutive 'not detected' results will remain within the analysis.

The time to confirmed negative test will be summarised descriptively by treatment group. Kaplan Meier [2] curves will be produced for each treatment group, overlayed on one plot. A supporting table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants without a negative test, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].

Time to Confirmed Negative Test by qRT-PCR Measurements in Nasal Samples Starting from Peak qRT-PCR after Initial Administration of IMP to First Confirmed Undetectable Assessment after Peak Measure

The time from the peak qRT-PCR measurement after administration of IMP to the first confirmed negative qRT-PCR test will be calculated in days as:

Date and time of first confirmed negative test – Date and time of first IMP administration.

A negative test is defined as two consecutive 'Not Detected' results in the qRT-PCR test, with the date and time of the first negative test being utilised in the calculations. The peak qRT-PCR is defined as the highest viral load value obtained by a participant after their first administration of IMP.

Participants who did not have a confirmed undetectable assessment after their peak qRT-PCR after first administration of IMP are censored at their last detectable assessment. Participants who stay undetectable during guarantine will be excluded from this analysis.

The time to confirmed negative test will be summarised descriptively by treatment group. Kaplan Meier curves will be produced for each treatment group, overlayed on one plot. A supporting table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants without a negative test, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].

# Time to Peak qRT-PCR in Nasal Samples Starting from Initial Administration of IMP

The time to the peak qRT-PCR measurement starting from the initial administration of IMP will be calculated in days as:

Date and time of peak qRT-PCR measurement – Date and time of first IMP administration.

The peak qRT-PCR measurement is defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who stay undetectable during quarantine will be excluded from this analysis.

The time to peak qRT-PCR measurement will be summarised descriptively by treatment group. Kaplan Meier curves will be produced for each treatment group, overlayed on one plot. A supporting table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants not yet reaching peak qRT-PCR, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].

Area under the Viral Load-Time Curve (VL-AUC) of RSV Challenge Virus as Determined by Viral Culture in Nasal Samples, Starting from Initial Administration of IMP up to Planned Discharge from Quarantine

The area under the viral-load curve (VL-AUC) for RSV-A Memphis 37b measured in nasal washes by viral culture, from the last measurement collected prior to the first dose of IMP until the morning of Day 12 (Quarantine discharge) will be summarised and analysed as described in Section 10.7.1.

Viral culture analysis is only carried out on samples where the qRT-PCR results is at least detectable. Any missing viral culture results will be imputed with 'Not Detected' if the corresponding qRT-PCR result is not detected.

Peak Viral Load of RSV as Defined by the Maximum Viral Load determined by Viral Culture Measurements in Nasal Samples Starting from Initial Administration of IMP up to Planned Discharge From Quarantine

Using the scheduled protocol assessments from the last measurement collected prior to the first dose of IMP to the morning of Day 12 (Quarantine discharge), the highest viral culture measurement observed in nasal samples for each participant will be summarised and analysed in a similar fashion to the primary efficacy endpoint described in Section 10.7.1.

Participants who stay undetectable (i.e. a 'Not Detected' value) during quarantine will be replaced with the 'Not Detected' value shown in the table in Appendix 15.1.

Time to Confirmed Negative Test by Viral Culture Measurements in Nasal Samples Starting from Initial Administration of IMP to First Confirmed Undetectable Assessment after Peak Measure

The time from the first administration of IMP to the first confirmed negative viral culture measurement after the peak viral culture measurement will be calculated in days as:

Date and time of first confirmed negative test after peak viral culture measurement – Date and time of first IMP administration.

A negative test is defined as a 'Not Detected' result in the viral culture test, with the date and time of the first negative test being utilised in the calculations. The peak viral culture measurement is defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who did not have a confirmed undetectable assessment after first administration of IMP are censored at their last detectable assessment after their peak viral culture measurement. Participants who stay undetectable during quarantine will be excluded from this analysis.

The time to the confirmed negative test will be summarised descriptively by treatment group. Kaplan Meier curves will be produced for each treatment group, overlayed on one plot. A supporting table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants without a negative test, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].

Time to Confirmed Negative Test by Viral Culture Measurements in Nasal Samples Starting from Peak Viral Culture after Initial Administration of IMP to First Confirmed Undetectable Assessment after Peak Measure

The time from the peak viral culture measurement after administration of IMP to the first confirmed negative viral culture measurement will be calculated in days as:

Date of and time first confirmed negative test – Date and time of first IMP administration.

A negative test is defined as two consecutive 'Not Detected' results in the viral culture test, with the date and time of the first negative test being utilised in the calculations. The peak viral culture measurement is defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who did not have a confirmed undetectable assessment after their peak viral culture measurement after first administration of IMP are censored at their last detectable assessment. Participants who stay undetectable during quarantine will be excluded from this analysis.

The time to confirmed negative test will be summarised descriptively by treatment group. Kaplan Meier curves will be produced for each treatment group, overlayed on one plot. A supporting table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants without a negative test, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].
## Time to Peak qRT-PCR in Nasal Samples Starting from Initial Administration of IMP

The time to the peak qRT-PCR measurement starting from the initial administration of IMP will be calculated in days as:

Date and time of peak qRT-PCR measurement – Date and time of first IMP administration.

The peak qRT-PCR measurement is defined as the highest viral load value obtained by a participant after their first administration of IMP. Participants who stay undetectable during quarantine will be excluded from this analysis.

The time to peak qRT-PCR measurement will be summarised using a descriptive summary. Kaplan Meier curves will be produced for each treatment group, overlayed on one plot. A supporting summary table will include the median, 25<sup>th</sup> and 75<sup>th</sup> percentiles for each group and will be accompanied by a log rank test to compare between RV299 and placebo with the corresponding p-value presented.

[Kaplan-Meier plot: y-axis = cumulative proportion of participants not yet reaching peak qRT-PCR, x-axis = day relative to initial administration of IMP, one line for each treatment overlayed on the same plot].

## 10.7.2.4 Clinical Symptom-Related Endpoints

Area under the Curve over Time of Total Clinical Symptoms (TSS-AUC) as Measured from 10 Symptoms within the Graded Symptom Scoring System Collected 3 Times Daily Starting at Initial Administration of IMP up to Planned Discharge from Quarantine

Total symptom scores (from 10 items of the 13-item symptom diary card) will be used to calculate the AUC, from the assessment nearest to the time of the first administration of IMP (can be prior to or after dosing, depending on whether dosed in the morning or evening), i.e. baseline, until Day 12 (Quarantine discharge), for each participant using the trapezoidal rule [1].

Symptoms are assessed 3 times daily for Day 1 to Day 11 (and once for Day 12) and recorded on the symptom diary cards at each assessment. The following types of symptoms are recorded (on a grading scale, 0 to 3 (or 0 to 4 for the Shortness of Breath symptom)):

- Upper Respiratory Tract (URT): runny nose, stuffy nose, sore throat, sneezing, earache.
- Lower Respiratory Tract (LRT): cough, shortness of breath.
- Systemic: headache, malaise, muscle/joint ache/stiffness.
- Not used for analyses: chilliness/feverishness, chest tightness, wheeze.

A total symptom score will be derived for each participant, separately for each assessment (symptom diary card) on each day (Day 0 to Day 12) as follows:

- For each assessment, sum the 10 observed symptom grade values for each symptom diary card to obtain a total symptom score for each symptom diary card. If the participant does not have all 10 observed values on a specific symptom diary card being considered, then total symptom score will not be calculated for that symptom diary card. It is expected that participants will not have missing data.
- The AUC calculation will be based on the available non-missing calculated total symptom scores between the start and end of the defined AUC time. However, for an AUC to be derived, the participant should have at least 1 non-missing calculated total symptom scores at the start of the AUC period (e.g. date of first dose of IMP) and also at the end of the AUC time period

(e.g. Day 12). In addition, the participant should have at least 2 non-missing data recording on each day between the day after the start, and the day before the end, of the defined AUC time period (i.e. at least 2 out of the 3 possible assessments on each Day)). Any missing total symptom score data will be reviewed at the BDRM, for its potential impact on this endpoint, and any decisions to exclude participants as a result of these criteria will be documented in the BDRM minutes.

 As symptoms are scheduled to be taken 3 times daily for Days 0 to 11 (and once on Day 12), in order to calculate the AUC, the actual time that the assessment was collected will be used within the AUC calculation starting from the assessment at the time of the first administration of IMP.

The AUC of the total symptom score will be summarised by treatment group and modelled in the same way as the main analysis of the primary endpoint described in Section 10.7.1, including sensitivity analyses 1 and 2, as described therein.

The total symptom scores and the change from baseline scores will be summarised by timepoint (i.e. day relative to first administration of IMP and assessment) and treatment group. The symptom scores and the visual analogue score (VAS) in millimetres from the 13-item symptom diary card will be listed.

As well as a descriptive statistics summary of total symptom score values, the mean total symptom score values (+/- 1 Standard Error (SE)) will be displayed graphically by day (relative to first dose of IMP) and assessment, and treatment group. In order to calculate the time point that each assessment will be presented against, a relative day and relative assessment will be assigned. The last total symptom score measurement collected at the time of the first dose of IMP will be assigned to be the value at time point 1, while measurements collected on subsequent assessments and days will be assigned to subsequent time points in sequential order (i.e. time point 2, 3 and so on). Time point 1 will be presented against Day 0 assessment 1, while subsequent time points will be presented against Day 0 assessment 2, Day 0 assessment 3, Day 1 assessment 1, and so on. Negative timepoints relative to dosing will also be included and will be presented as Day -1 assessment 1.

[Line graph: y-axis = mean of total symptoms score, x-axis = day relative to dosing (the axis will be negative to include days prior to IMP administration), one line for each treatment group on same plot].

A boxplot will also be presented by day (relative to first dose of IMP) and assessment, plotting the median and mean qRT-PCT values for each treatment group, with the corresponding summary statistics.

[Box plot: y-axis = mean of qRT-PCR ( $log_{10}$  copies/mL), x-axis = day relative to dosing, one box-and-whisker for each day, with each treatment panelled with RV299 at the top and placebo below].

Note: For multiple assessments taken within each day, so as to be able to plot mean values across participants (within a treatment group) by day, the actual collection time point (which may differ across participants) will not be used. Rather all first, second and third assessments will have mean values separately calculated and plotted as three means within each day. These three means will be shown equally spaced along the x-axis within the graph.

Area under the Curve over Time of Total Clinical Symptoms Change from Baseline (TSS-AUC-CFB) as Measured from 10 Symptoms within the Graded Symptom Scoring System Collected 3 Times Daily Starting at Initial Administration of IMP up to Planned Discharge from Quarantine

The change from baseline will be calculated for each assessment following administration of IMP and an AUC calculated using these scores will be analysed in the same manner as described above

(including sensitivity analyses 1 and 2), where the baseline assessment is the assessment nearest to the time of the first administration of IMP (can be prior to or after dosing, depending on whether dosed in the morning or evening).

Peak Symptoms Diary Card Score: Peak Total Clinical Symptoms (TSS) as Measured from 10 Symptoms within the Graded Symptom Scoring System Collected 3 Times Daily Starting from Initial Administration of IMP up to Planned Discharge from Quarantine

Using the scheduled protocol assessments from the assessment at the time of the first dose of IMP to Day 12 (Quarantine discharge), the highest total symptom score (defined as the sum of all 10 individual composite symptoms) will be summarised by treatment group and modelled in the same way as the main analysis of the primary endpoint.

Participants who do not record any symptoms will be assigned a peak of 0.

Peak Daily Symptom Score: Individual Maximum Daily Sum of Symptom Score from Initial Administration of IMP up to Planned Discharge from Quarantine

The highest total symptom score recorded on each day, across the three assessments, for each participant will be summarised descriptively by treatment group and assessment day.

Time to Symptom Resolution as Measured from 10 Symptoms within the Graded Daily Symptom Scoring System Starting at Initial Administration of IMP to 24-hours Symptom Free

Symptom resolution is defined as a participant scoring 0 for the total symptom score for a 24 hour period (e.g a minimum of three consecutive symptom diary cards, each with a score of 0) after their peak symptom score.

The time from the assessment at the time of the first administration of IMP until symptom resolution will be calculated in days as:

Date and time of symptom resolution – Date and time of assessment at IMP administration.

The time to symptom resolution will be summarised by treatment group using descriptive summaries.

If the peak symptom score occurs on more than one day then the first occurrence will be selected. Participants who do not record 24 hours symptom free after their highest total symptom score during the quarantine period will be censored at their last assessment and participants who record no symptoms during quarantine will be excluded from this analysis.

Time to Symptom Resolution as Measured from 10 Symptoms within the Graded Daily Symptom Scoring System Starting at Peak Symptoms after Initial Administration of IMP to 24-hours Symptom

The time from the highest total symptom score following administration of IMP until symptom resolution will be calculated in days as:

Date and time of symptom resolution – Date and time of highest total symptom score.

The time to symptom resolution after the peak symptom score will be summarised by treatment group using descriptive summaries.

If the peak symptom score occurs on more than one day then the first occurrence will be selected. Participants who do not record 24 hours symptom free after their highest total symptom score during the quarantine period will be censored at their last assessment and participants who record no symptoms during quarantine will excluded from this analysis.

# Time to Peak as Measured from 10 Symptoms within the Graded Daily Symptom Scoring System Starting from Initial Administration of IMP to the Time of Peak Daily Symptom Score

The time from the assessment at the time of the first dose of IMP (can be prior to or after dosing, depending on whether dosed in the morning or evening) until the highest total symptom score will be calculated in days as:

Date and time of highest total symptom score – Date of and time of assessment at IMP administration.

The time to peak daily symptom score will be summarised by treatment group using descriptive summaries.

If the peak symptom score occurs on more than one day then the first occurrence will be selected. Participants who record no symptoms during quarantine will be censored at their last assessment.

## 10.7.2.5 Nasal Discharge Endpoints

## Total Weight of Mucus Produced Starting at Initial Administration of IMP up to Planned Discharge from Quarantine

Total weight of nasal mucus (grams) will be calculated as the sum of mucus weights taken from the assessment at the time of the first administration of IMP (can be prior to or after dosing, depending on whether dosed in the morning or evening) to morning of Day 12 (Quarantine discharge). Total mucus weight will be summarised by treatment group and will include the change from baseline, where baseline is the last assessment recorded prior to receiving a positive result for RSV by qicPCR. For participants who did not receive a positive result, the final assessment prior to the first administration of IMP will be defined as the baseline score.

# Total Number of Tissues Used by Participants Starting At Initial Administration of IMP up to Planned Discharge from Quarantine

Total number of tissues will be counted from the assessment at the time of the first dose of IMP (can be prior to or after dosing, depending on whether dosed in the morning or evening) to morning of Day 12 (Quarantine discharge). This count will be summarised by treatment group and will include the change from baseline, where baseline is the last assessment recorded prior to receiving a positive result for RSV by qicPCR. For participants who did not receive a positive result, the final assessment prior to the first administration of IMP will be defined as the baseline score.



| CCI |
|-----|
| CCI |



## 10.8. Pharmacokinetic Analysis

Summary of the pharmacokinetic (PK) data and endpoints will not be performed by S-cubed and will therefore not be a part of this SAP. Details of the PK Analysis will be found in the CPAP provided by VENN. Discussion of the PK parameter correlation can be found in Section 10.7.3.1..

## 10.9. Safety Analysis

All analyses of safety endpoints will be descriptive only. The safety population will be used for all safety presentations.

#### 10.9.1. Adverse Events

All adverse events (AE) will be coded using MedDRA, Version 25.0.

An adverse event is defined as treatment emergent if the onset date is on or after the date of first dosing with IMP. Should any onset date for an adverse event be missing or only a partial date recorded (such that it cannot be determined if the event onset was prior to start of IMP or not) then it will be assumed that the event is treatment emergent, unless the adverse event stop date indicates otherwise.

Similarly, an AE is defined as challenge emergent if the onset date is on or after the date of inoculation. Should any onset date for an adverse event be missing or only a partial date recorded (such that it cannot be determined if the event onset was prior to inoculation or not) then it will be assumed that the event is challenge emergent, unless the adverse event stop date indicates otherwise.

An AE can be both challenge emergent and treatment emergent. Any AE with an onset date earlier than the inoculation date will be classified as a pre-treatment AE.

If a participant experiences more than one adverse event with the same preferred term, that preferred term will be counted only once. It will be assigned the greatest observed severity and the strongest relationship to IMP among those events for the tables in which those characteristics are summarised.

Pre-treatment AEs will be identified in a patient listing.

A summary of treatment-emergent AEs will be presented by treatment group showing the number of events, number of participants with events (also split by severity; mild, moderate, severe), number of participants with SAEs, number of participants with related events, number of participants with events

leading to early withdrawal from the study and the number of participants with events leading to early discontinuation of IMP.

Further summaries will present the treatment-emergent AEs by:

- Treatment group, SOC and PT.
- Treatment group, SOC, PT and severity.
- Treatment group, SOC, PT and relationship to IMP.

Further summaries will present the challenge-emergent AEs by:

• Treatment group, SOC, PT and relationship to challenge agent.

Tables presented by relationship will only include the subset of adverse events that are judged as being 'Related' to IMP or challenge agent, i.e. correspond to adverse events where relationship is recorded on the adverse event page as being 'Unlikely', 'Possibly', 'Probably', 'Definitely', or a relationship is not given.

In all AE summary tables results will be displayed ordered in terms of decreasing frequency of SOC occurrence (based on total across all participants), and within each SOC also ordered in terms of decreasing frequency of preferred term occurrence (also based on total across all participants). In all AE summary tables a total column including data across all participants will also be presented.

## 10.9.2. Laboratory Variables

For all laboratory variables, baseline is defined as the assessment collected prior to the first administration of IMP.

The following parameters will be included within summary presentations (and presented in the units as shown):

- Haematology: platelet count (10^9/L), white blood cell (WBC) count (absolute) (10^9/L), neutrophils (% and absolute (10^9/L)), lymphocytes (% and absolute (10^9/L)), monocytes (% and absolute (10^9/L)), eosinophils (% and absolute (10^9/L)), basophils (% and absolute (10^9/L)), red blood cell (RBC) count (10^12/L), reticulocyte count (% and absolute (10^9/L), haemoglobin (g/L), haematocrit (%), mean corpuscular volume (MCV) (fL), mean corpuscular haemoglobin (MCH) (PG), mean corpuscular haemoglobin concentration (MCHC) (g/L).
- Coagulation: prothrombin time (PT) (secs), activated partial thromboplastin time (APTT) (secs).
- Biochemistry: sodium (mmol/L), potassium (mmol/L), glucose (mmol/L), albumin (g/L), chloride (mmol/L), bicarbonate (mmol/L), calcium (mmol/L), uric acid (umol/L), total protein (g/L), creatinine (umol/L), total bilirubin (umol/L), indirect bilirubin (umol/L), direct bilirubin (umol/L), inorganic phosphate (mmol/L), blood urea nitrogen (mg/dL), C-reactive protein (CRP) (mg/L), gamma glutamyl transferase (GGT) (IU/L), alkaline phosphatase (ALP) (IU/L), alanine transaminase (ALT) (IU/L), lactate dehydrogenase (LDH) (IU/L), aspartate transaminase (AST) (IU/L), urea (mmol/L).
- Thyroid Function Tests (screening only): Free thyroxine (pmol/L), Thyroid Stimulating Hormone (mIU/L).
- Cardiac Enzymes: creatine kinase (IU/L), troponin T (ng/L).
- Urinalysis: colour, specific gravity, appearance, pH, dipstick presence of: blood, glucose, leukocytes, ketones, nitrite, protein, urobilinogen, bilirubin.

• Human Immunodeficiency Virus and Hepatitis A, B and C: HIV-1 and HIV-2 antibodies, hepatitis A antibodies (HepA IgM), hepatitis B surface antigen (HBsAg), hepatitis C antibodies (HCAb).

Observed parameter values and changes from baseline will be summarised appropriately for the above haematology, chemistry, coagulation and cardiac enzyme parameters. Any other laboratory parameters collected as part of the study will only be included in participant listings. Laboratory data collected in different units to that shown will be converted to the above specified units (if possible) for presentation in tables and listings.

Laboratory values outside the reference range will be identified in the participant listings as above or below the reference range. Laboratory values that are below the limit of quantification (BLQ) will be set to zero in computations for summary presentations but will be noted as BLQ in participant listings. Laboratory values that are missing will remain missing and will be noted as such in listings.

## 10.9.3. Vital Signs

Vital signs parameters to be summarised are:

 Heart Rate (beats per minute), systolic blood pressure (mmHg), diastolic blood pressure (mmHg), respiratory rate (breaths per minute), peripheral arterial oxygen saturation (%) and tympanic temperature (°C).

Vital signs parameters will be summarised as observed parameter values and changes from baseline, by treatment group for all scheduled protocol visits, where baseline is defined as the assessment performed prior to the first administration of IMP.

## 10.9.4. Spirometry

Summary statistics for absolute values and change from baseline by time point will be tabulated, by group, for spirometry parameters (FEV<sub>1</sub>(absolute), FEV<sub>1</sub>(% predicted), Forced vital capacity (FVC) (absolute), FVC (% predicted), FEV<sub>1</sub>/FVC ratio (absolute), FEV<sub>1</sub>/FVC ratio (% predicted)) and will also be included within participant listings.

The spirometry baseline is the assessment performed at screening.

## **10.9.5.** Physical Examination

Physical examination findings (both for the complete examination and also any directed examination assessments) will be included within participant listings.

## 10.9.6. 12-Lead Electrocardiograms

Summary statistics for absolute values and change from baseline by time point will be tabulated, by treatment group for the following ECG parameters: (Heart Rate (bpm), PR interval (sec), QRS duration (sec), QT interval (sec), QTc interval (sec), QTcB interval (sec), QTcF interval (sec) and RR interval (sec)). For all ECG parameters, the baseline assessment is defined as the assessment performed prior to IMP dosing. All data will be included within participant listings.

# 11. CHANGES TO THE PROTOCOL SPECIFIED ANALYSIS DETAILED IN THE STATISTICAL ANALYSIS PLAN

- 1. Clarity has been added to the definitions for the ITT-A and ITT-B populations to ensure they are mutually exclusive and are accounting for subjects who have a positive detection either side of IMP administration.
- 2. The protocol incorrectly used median AUC as the main estimator of the primary endpoint. This has been corrected within the SAP to use the mean AUC.
- 3. Inferential analysis was not required for any time to event secondary endpoints within the protocol. However, this have been deemed as necessary to support the study outcome and log rank tests have been added to the appropriate endpoints.
- 4. The endpoint 'Time (days) to peak viral culture in nasal samples, starting from initial administration of IMP' had been missed in the list of endpoints within the protocol, though referred to in later sections. This endpoint has been added to the SAP.
- 5. Symptom resolution was included within the wording of the secondary clinical-symptom related endpoints and referred to as 'returning to baseline score'. This was deemed not to fit the requirements of the endpoint and has instead been amended to be 24-hours symptom free.
- 6. The endpoint 'Time to symptom resolution ... starting at initial administration of IMP to time of returning to baseline score' has been expanded to include the caveat that the symptom-free period must occur after the peak symptom score.

## 12. REFERENCES

[1] Matthews JNS, Altman DG, Campbell MJ, Royston P. Analysis of serial measurements in medical research. *Br Med J* (1990); 300: 230-5.

[2] Kaplan EL, Meier P. Nonparametric estimation from incomplete observations. Journal of American Statistical Association. 1958; 53:457-481.

## 13. TABLES, FIGURES AND LISTINGS

## 13.1. Specific Presentation Details

Tables, listings, and figures will be provided in a WORD document [and programmed off CDISC compliant SDTM SAS data sets.]. All summary tables and figures will have source data footnotes that refer to the relevant listings. Dates will appear as ddmmmyyyy; times as hh:mm. All listings will be ordered by treatment group, participant number, and scheduled visit. For the presentation of summary data, values will be aligned based on the unit column, and not left/right justified. For example:

| Parameter | n | xx | XX |
|-----------|-----------|--------------|--------------|
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | GM (GSD) | xx.x (xx.xx) | xx.x (xx.xx) |
| | %CV | XX.X | XX.X |
| | SE | xx.xx | XX.XX |
| | Median | xx.x | XX.X |
| | Q1, Q3 | XX.X, XX.X | XX.X, XX.X |
| | Min, Max | XX, XX | xx, xx |

All tables, listings and figures will have the SAS program name, output filename and date of production in the footnote.

All tables, listings and figures will include the following study header and footer:

CONFIDENTIAL hVIVO Services Ltd Page x of y REVD002 [VIR-CST-001]

Table x.x Title Participant population

Source Data: Listing 16.2.x {Source data footnote only appears for tables, where x references relevant listing number}

Program: xxxxxxxxx Output: xxxxxxxx Date: xxxxxxxxx

#### 13.2. List of Tables

For the primary endpoint and selected secondary occurrence tables will be repeated for the ITT-A, ITT-B, ITT and PP Populations where the difference between the ITT-I is greater than 1 participant within a treatment group. Where tables are to be repeated on any additional populations, an X has been marked in the relevant column. If a table is repeated, the original table number as produced for the ITT-I population will have .1 added and this final digit will be increased by 1 for repeats on the ITT-A. Similarly, for repeats on ITT-B the number will increase by 2, for repeats on ITT the number will increase by 3 and for repeats on the PP the number will increase by 4. For example, table 14.2.1.1 will be produced for the ITT-I population and will be repeated as 14.2.1.2, 14.2.1.3, 14.2.1.4 and 14.2.1.5 for the ITT-A, ITT-B, ITT and PP populations respectively. If no repeats of a table are required then the original table will not require the final .1.

| | | Repeated for | | | |
|---|---|---|---|---|---|
| Table<br>Number | Table Title | ITT-<br>A | ITT-<br>B | ITT | PP |
| 14.1.1 | Participant Disposition – All Participants | | | | |
| 14.1.2 | Demography – Safety Population | | | | |
| 14.1.3 | IMP Exposure and Compliance – Safety Population | | | | |
| 14.1.4 | Concomitant Medications – Safety Population | | | | |
| 14.2.1.1 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Initial Administration of IMP to Quarantine Discharge – ITT-I Population | X | X | X | X |
| 14.2.1.2 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Initial Administration of IMP for 6.5 Days – ITT-I Population | Χ | | | |
| 14.2.1.3 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Day 2 to Day 12 – ITT-I Population | Χ | | | |
| 14.2.1.4 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Initial Administration of IMP to Quarantine Discharge (Untransformed Data) – ITT-I Population | X | | | |
| 14.2.2.1 | Peak Viral Load of RSV Challenge Virus by qRT-PCR from Initial Administration of IMP to Quarantine Discharge – ITT-I Population | X | | | |
| 14.2.2.2 | Time to First Confirmed Undetectable Assessment of RSV Challenge Virus by qRT-PCR from Initial Administration of IMP – ITT-I Population | X | | | |
| 14.2.2.3 | Time to First Confirmed Undetectable Assessment of RSV Challenge Virus after Peak Measure by qRT-PCR following Initial Administration of IMP – ITT-I Population | X | | | |
| 14.2.2.4 | Time to Peak RSV Challenge Virus by qRT-PCR following Initial Administration of IMP – ITT-I Population | Χ | | | |
| 14.2.2.5.1 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP to Quarantine Discharge – ITT-I Population | X | Х | X | Х |
| 14.2.2.5.2 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP for 6.5 Days – ITT-I Population | Χ | | | |
| 14.2.2.5.3 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Day 2 to Day 12 – ITT-I Population | X | | | |

| Table | | - | Repeated for ITT- ITT | | |
|---|---|---|---|---|---|
| Number | Table Title | Α | В | "" | PP |
| 14.2.2.5.4 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP to Quarantine Discharge (Untransformed Data) – ITT-I Population | Х | | | |
| 14.2.2.6 | Peak Viral Load of RSV Challenge Virus by Viral Culture from Initial Administration of IMP to Quarantine Discharge – ITT-I Population | X | | | |
| 14.2.2.7 | Time to First Confirmed Undetectable Assessment of RSV Challenge Virus after Peak Measure by Viral Culture starting from Initial Administration of IMP - ITT-I Population | X | | | |
| 14.2.2.8 | Time to First Confirmed Undetectable Assessment of RSV Challenge Virus by Viral Culture starting from Peak Measure - ITT-I Population | X | | | |
| 14.2.2.9 | Time to Peak RSV Challenge Virus by Viral Culture following Initial Administration of IMP – ITT-I Population | Х | | | |
| 14.2.3.1.1 | AUC of Total Symptom Score from 10-Item Diary Card from First Administration of IMP to Quarantine Discharge - ITT-I Population | X | X | X | X |
| 14.2.3.1.2 | AUC of Total Symptom Score from 10-Item Diary Card from First Administration of IMP for 6.5 Days - ITT-I Population | Χ | | | |
| 14.2.3.1.3 | AUC of Total Symptom Score from 10-Item Diary Card from Day 2 to Day 12 - ITT-I Population | Χ | | | |
| 14.2.3.2.1 | AUC of Total Symptom Score Change from Baseline from 10-<br>Item Diary Card from First Administration of IMP to<br>Quarantine Discharge - ITT-I Population | X | X | X | X |
| 14.2.3.2.2 | AUC of Total Symptom Score Change from Baseline from 10-<br>Item Diary Card from First Administration of IMP for 6.5 days<br>- ITT-I Population | X | | | |
| 14.2.3.2.3 | AUC of Total Symptom Score Change from Baseline from 10-<br>Item Diary Card from Day 2 to Day 12 - ITT-I Population | X | | | |
| 14.2.3.3 | Total Symptom Score from 10-Item Diary Card by Assessment - ITT-I Population | Χ | Χ | X | Χ |
| 14.2.3.4 | Peak Total Symptom Score from 10-Item Diary Card from First Administration of IMP to Quarantine Discharge - ITT-I Population | X | | | |
| 14.2.3.5 | Peak Total Symptom Score from 10-Item Diary Card by Day - ITT-I Population | | | | |
| 14.2.3.6 | Peak Daily Symptom Score from 10-Item Diary Card - ITT-I<br>Population | | | | |
| 14.2.3.7 | Time to Symptom Resolution by 10-Item Diary Card from Initial Administration of IMP to 24-Hours Symptom Free - ITT-I Population | X | | | |
| 14.2.3.8 | Time to Symptom Resolution by 10-Item Diary Card from Peak Total Symptom Score to 24-Hours Symptom Free - ITT-I Population | X | | | |

| | | - | eated f | or | |
|---|---|---|---|---|---|
| Table<br>Number | Table Title | ITT- | ITT-<br>B | IΠ | PP |
| 14.2.3.9 | Time to Peak Symptom Score by 10-Item Diary Card from | X | В | | |
| 14.2.3.3 | Initial Administration of IMP - ITT-I Population | ^ | | | |
| 14.2.4.1 | Total Weight of Mucus Produced from Initial Administration of IMP to Quarantine Discharge by Assessment - ITT-I Population | X | | | |
| 14.2.4.2 | Total Number of Tissues Used from Initial Administration of IMP to Quarantine Discharge by Assessment - ITT-I Population | | | | |
| CCI | | | | | |
| | | X | | | |
| | | ^ | | | |
| 14.3.1.1 | Overall Summary of Treatment Emergent Adverse Events – Safety Population | | | | |
| 14.3.1.2 | Treatment Emergent Adverse Events by System Organ Class and Preferred Term – Safety Population | | | | |
| 14.3.1.3 | Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Severity – Safety Population | | | | |
| 14.3.1.4 | Treatment Emergent Adverse Events Related to RV299 by System Organ Class and Preferred Term— Safety Population | | | | |
| 14.3.1.5 | Adverse Events Related to Challenge Agent by System Organ<br>Class and Preferred Term – Safety Population | | | | |
| 14.3.2 | Haematology Parameters: Summary – Safety Population | | | | |
| 14.3.3 | Biochemistry Parameters: Summary – Safety Population | | | | |
| 14.3.4 | Coagulation Parameters: Summary – Safety Population | | | | |
| 14.3.5 | Cardiac Enzymes Parameters: Summary – Safety Population | | | | |
| 14.3.6 | Urinalysis Parameters: Summary – Safety Population | | | | |
| 14.3.7 | Vital Signs Parameters: Summary – Safety Population | | | | |
| 14.3.8 | Spirometry Parameters: Summary – Safety Population | | | | |
| 14.3.9 | 12-Lead Electrocardiogram Parameters: Summary – Safety Population | | | | |

## 13.3. List of Figures

For the primary endpoint and selected secondary CGI figures will be repeated for the ITT-A, ITT-B, ITT and PP Populations where the difference between the ITT-I is greater than 1 participant within a treatment group. Where figures are to be repeated on any additional populations, an X has been marked in the relevant column. If a figure is repeated, the original figure number as produced for the ITT-I population will have .1 added and this final digit will be increased by 1 for repeats on the ITT-A. Similarly, for repeats on ITT-B the number will increase by 2, for repeats on ITT the number will increase by 3 and for repeats on the PP the number will increase by 4. For example, figure 14.2.1.1 will be produced for the ITT-I population and will be repeated as 14.2.1.2, 14.2.1.3, 14.2.1.4 and 14.2.1.5 for the ITT-A, ITT-B, ITT and PP populations respectively. If no repeats of a table are required then the original table will not require the final .1.

| | ten the original table will not require the mar.1. | Repe | ated f | or | |
|---|---|---|---|---|---|
| Figure<br>Number | Figure Title | ITT-<br>A | ITT-<br>B | ITT | PP |
| 14.2.1.1 | Mean RSV Challenge Virus Viral Load by qRT-PCR by Days from IMP Administration – ITT-I Population | Χ | X | Χ | X |
| 14.2.1.2 | Boxplot of RSV Challenge Virus Viral Load by qRT-PCR by Days from IMP Administration – ITT-I Population | Χ | X | Χ | Х |
| 14.2.2.1 | Peak RSV Challenge Virus Viral Load by qRT-PCR by Days from IMP Administration – ITT-I Population | X | | | |
| 14.2.2.2 | Kaplan-Meier Plot of Time to First Confirmed Undetectable<br>Assessment of RSV Challenge Virus by qRT-PCR from Initial<br>Administration of IMP – ITT-I Analysis Set | Х | | | |
| 14.2.2.3 | Kaplan-Meier Plot of Time to First Confirmed Undetectable<br>Assessment of RSV Challenge Virus after Peak Measure by<br>qRT-PCR following Initial Administration of IMP – ITT-I<br>Population | X | | | |
| 14.2.2.4 | Kaplan-Meier Plot of Time to Peak RSV Challenge Virus by qRT-PCR following Initial Administration of IMP — ITT-I Population | X | | | |
| 14.2.2.5.1 | Mean RSV Challenge Virus Viral Load by Viral Culture by Days from IMP Administration – ITT-I Population | Χ | X | Χ | Х |
| 14.2.2.5.2 | Boxplot of RSV Challenge Virus Viral Load by Viral Culture by Days from IMP Administration – ITT-I Population | X | X | Χ | Х |
| 14.2.2.6 | Peak RSV Challenge Virus Viral Load by Viral Culture by Days from IMP Administration – ITT-I Population | Х | | | |
| 14.2.2.7 | Kaplan-Meier Plot of First Confirmed Undetectable Assessment of RSV Challenge Virus after Peak Measure by Viral Culture starting from Initial Administration of IMP – ITT-I Population | X | | | |
| 14.2.2.8 | Kaplan-Meier Plot of First Confirmed Undetectable<br>Assessment of RSV Challenge Virus by Viral Culture starting<br>from Peak Measure – ITT-I Population | X | | | |
| 14.2.3.1.1 | Mean Daily Total Symptom Score from 10-item Diary Card by Days from IMP Administration – ITT-I Population | Χ | Х | Χ | Х |
| 14.2.3.2.1 | Peak Daily Total Symptom Score from 10-item Diary Card by Days from IMP Administration — ITT-I Population | X | | | |
| CCI | | | | | |

| | _ | Repe | eated f | or | |
|--------|--------------|------|---------|-----|----|
| Figure | | ITT- | | ITT | PP |
| Number | Figure Title | Α | В | | |
| CCI | | | | | |
| | | _ | | | |
| | | _ | | | |
| | | _ | | | |

## 13.4. List of Listings

| Listing Number | Listing Title |
|---|---|
| 16.2.1.1 | Participant Disposition |
| 16.2.1.2 | Failed Inclusion and Exclusion Criteria |
| 16.2.2 | Protocol Deviations |
| 16.2.3 | Participant Populations |
| 16.2.4.1 | Demographics |
| 16.2.4.2 | Reproductive Status and Contraceptive Use |
| 16.2.4.3 | Smoking History |
| 16.2.4.4 | Alcohol Use |
| 16.2.4.5 | Recreational Drugs of Abuse |
| 16.2.4.6 | Medical History |
| 16.2.4.7 | Prior and Concomitant Medications |
| 16.2.5.1 | Challenge Virus Inoculation Administration |
| 16.2.5.2 | Viral Shedding Results |
| 16.2.5.3 | IMP Administration |
| 16.2.6.1.1 | Viral Load by Nasal Samples qRT-PCR Results |
| 16.2.6.1.2 | Viral Load by Nasal Samples qRT-PCR Derivations |
| 16.2.6.2.1 | Viral Load by Nasal Samples Viral Culture Results |
| 16.2.6.2.2 | Viral Load by Nasal Samples Viral Culture Derivations |
| 16.2.6.3.1 | Symptom Scores from Symptom Diary Card |
| 16.2.6.3.2 | Visual Analogue Scale from Symptom Diary Card |
| 16.2.6.3.3 | Total Symptom Score: AUC Derivations |
| 16.2.6.3.4 | Total Symptom Score: Other Derivations |
| 16.2.6.4 | Mucus Weight and Tissue Bag Distribution |
| 16.2.6.5 | Nasopharyngeal Swab: Respiratory Virus Screen/Rapid Viral Antigen Test |
| 16.2.6.6 | Plasma PK Parameters |
| 16.2.7 | Adverse Events |
| 16.2.8.1 | Blood Sample Collection |
| 16.2.8.2 | Haematology |
| 16.2.8.3 | Coagulation |
| 16.2.8.4 | Biochemistry |
| 16.2.8.5 | Thyroid Function Tests |
| 16.2.8.6 | Cardiac Enzymes |
| 16.2.8.7 | Human Immunodeficiency Virus and Hepatitis A, B and C |
| 16.2.8.8.1 | Other Laboratory Tests: TDL |
| 16.2.8.9.1 | Other Laboratory Tests: Urine Pregnancy |
| 16.2.8.9.2 | Other Laboratory Tests: Drugs of Abuse Screen |
| 16.2.8.9.3 | Other Laboratory Tests: Urine Cotinine |
| 16.2.8.9.4 | Other Laboratory Tests: Alcohol Breath Test |
| 16.2.9.1 | Urinalysis |
| 16.2.9.2 | Urinalysis (TDL): Microscopy |

| Listing Number | Listing Title |
|----------------|-------------------------|
| 16.2.10 | Vital Signs |
| 16.2.11 | Spirometry |
| 16.2.12.1 | Physical Examination |
| 16.2.12.2 | Rhinoscopic Examination |
| 16.2.13 | ECG |
| 16.2.14 | Visit Dates |

## 14. TABLE AND LISTING SHELLS

Table 14.1.56
Participant Disposition
All Participants

| | | Treatme: | | | | |
|---|---|---|---|---|---|---|
| | | RV299 | Placebo | | | erall |
| | | (N=xx) | , | I=xx) | (N=xx) | |
| | n | (%) | n | (%) | n | (%) |
| Enrolled | | | | | XX | |
| Received challenge agent | | | | | XX | |
| Randomised | XX | | XX | | XX | |
| Received at least 1 dose of IMP | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Received all doses of IMP | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Received all doses of the | 2121 | (222.21) | 7171 | (1121.21) | 7171 | (2121 • 21) |
| ITT Population [1] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| ITT-I Population [2] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| ITT-A Population [3] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| ITT-B Population [4] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Per Protocol Population [5] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Safety Population [6] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X |
| PK Population [7] | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Discontinued IMP | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Completed study | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Withdrew from study | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Reason for Discontinuation of IMP: | | | | | | |
| Death | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Adverse Event | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Withdrawal by Subject | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Investigator's Decision | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Reason for Study Withdrawal: | | | | | | |
| Death | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Adverse Event | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Withdrawal by Subject | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Investigator's Decision | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Non-compliance with Study Requirements | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Pregnancy | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Study Terminated by Sponsor | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Lost to Follow-up | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Never dosed | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Other | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |

<sup>[1]</sup> Intent to Treat (ITT) Population = All randomised participants receiving challenge virus and at least one dose of IMP.

Note: Percentages are based on all randomised participants.

<sup>[2]</sup> Intent to Treat Infected (ITT-I) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection.

<sup>[3]</sup> Intent to Treat Infected Pre-dose (ITT-A) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection, using only assessments prior to taking IMP.

<sup>[4]</sup> Intent to Treat Infected Post-dose (ITT-B) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection, using only assessments after IMP.

<sup>[5]</sup> Per Protocol (PP) Population = All ITT-I population participants who have no major protocol deviations, and who complete the quarantine period up to the final day of quarantine (Study Day 12) and receive all 10 doses of IMP.

<sup>[6]</sup> Safety Population = All randomised participants receiving challenge virus and at least one dose of IMP.

<sup>[7]</sup> The PK Population = All ITT participants with at least one post-dose PK result.

<sup>[8]</sup> Completed Study = Participating in the study up to and including Day 28 (Follow-up).

Table 14.1.2 Demography Safety Population

| | | Treatment | Group | |
|---|---|---|---|---|
| | | RV299<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
| Ethnicity<br>Hispanic or Latino | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | | · | | |
| Not Hispanic or Latino | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Not Reported | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Unknown | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Race | | | | |
| American Indian or Alaska Native | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Asian | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Black or African American | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Native Hawaiian or Other Pacific Islander | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| White | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Other | n (%) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Height at Screening (m) | n | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| Weight at Screening (kg) | n | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX |
| | Min, Max | XX, XX | XX, XX | XX, XX |
| | MIII, Max | AA, AA | ΔΛ, ΔΛ | ^^, ^^ |
| BMI at Screening (kg/m^2) | n | XX | XX | XX |
| | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) |
| | Median | XX.X | XX.X | XX.X |
| | 01, 03 | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX |
| | Min, Max | XX, XX | XX, XX | XX, XX |

BMI = Body Mass Index

Note: Percentages are based on the safety population.

Programming note: If any categorical parameters have missing values for certain participants, then include a missing value category.

Table 14.1.3
IMP Exposure and Compliance
Safety Population

| | Treatment Group | | | |
|---|---|---|---|---|
| | | RV299<br>(N=xx) | Placebo<br>(N=xx) | Overall<br>(N=xx) |
| Number of doses of IMP received | n<br>Mean (SD)<br>Median<br>Q1, Q3<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, X.XX<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, X.XX<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X, X.XX<br>XX, XX |
| Compliance<br><80%<br>80% - 120%<br>>120% | n (%)<br>n (%)<br>n (%) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) | XX (XX.X)<br>XX (XX.X)<br>XX (XX.X) |

Note: Compliance = (number of doses received / number of doses expected) \* 100.

Table 14.1.4 Concomitant Medications Safety Population

| | | Treatme | nt Group | | | |
|---|---|---|---|---|---|---|
| Drug Class (L2)/ | | V299 | Place | | | rall |
| WHO Drug Name [1] | (N=xx) | | (N=xx) | | (N=xx) | |
| | n | % | n | % | n | જ |
| Number of Subjects with any Medication | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Drug Class 1 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| WHO Drug Name 1 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| WHO Drug Name 2 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Drug Class 2 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| WHO Drug Name 1 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| WHO Drug Name 2 | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |

<sup>[1]</sup> All medications will be coded using the WHO Drug Global Version March 1 2022.

Note: Concomitant medications correspond to medications where medication stop date is not before the date of IMP treatment.

Note: Table shows distinct number of participants with each WHO Drug Name/Drug Class.

| | Treatmen | nt Group |
|----------------------------------------|----------------|--------------|
| AUC(hours*Log10 copies/mL) | RV299 | Placebo |
| | (N=xx) | (N=xx) |
| n | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| %CV | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, X.XX | XX.X, X.XX |
| Min, Max | XX, XX | XX, XX |
| Difference in LS means [1] | XX.XX | |
| 95% Confidence interval for difference | XX.XXX, XX.XXX | |
| P-value [1] | X.XXX | |

[1] Comparison of RV299 and placebo using an ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate.

This table may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

This layout will be utilised for the following tables:

| Table 14.2.1.2 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Initial Administration of IMP for 6.5 Days - ITT-I Population |
|---|---|
| Table 14.2.1.3 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Day 2 to Day 12 - ITT-I Population |
| Table 14.2.1.4 | AUC of RSV Challenge Virus Viral Load by qRT-PCR from Initial Administration of IMP to Quarantine Discharge (Untransformed Data) - ITT-I Population |
| Table 14.2.2.1 | Peak Viral Load of RSV Challenge Virus by qRT-PCR from Initial Administration of IMP to Quarantine Discharge - ITT-I Population |
| | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP to Quarantine Discharge - ITT-I Population |
| Table 14.2.2.5.2 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP for 6.5 Days - ITT-I Population |
| | AUC of RSV Challenge Virus Viral Load by Viral Culture from Day 2 to Day 12 - ITT-I Population |
| Table 14.2.2.5.4 | AUC of RSV Challenge Virus Viral Load by Viral Culture from Initial Administration of IMP to Quarantine Discharge (Untransformed Data) - ITT-I Population |
| Table 14.2.2.6 | Peak Viral Load of RSV Challenge Virus by Viral Culture from Initial Administration of IMP to Quarantine Discharge - ITT-I Population |

Where appropriate, these tables may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

Programming Note: It is possible that the parametric methods will fail to meet the required assumptions for the main or repeated tables. Therefore, we will provide a Wilcoxon test (see Section 10.1.4). The alternative presentation for this is shown below and will require the following footnote to be updated: [1] Comparison of RV299 and placebo using a Wilcoxon rank sum test.

Version 01-00, 20DEC2022

Median difference in LS means [1] XX.XX P-value [1] X.XXX

 ${\it Table 14.2.2.2.1}$  Time to First Confirmed Undetectable Assessment of RSV Challenge Virus by qRT-PCR from Initial Administration of IMP ITT-I Population

| | | | Treatme | nt Group | | |
|---|---|---|---|---|---|---|
| | | RV299<br>(N=xx) | | | Placeb<br>(N=xxx | |
| | | | Kaplan-Meier | | | Kaplan-Meier |
| ime (days) | n | N# | Estimate | n | N# | Estimate |
| X | xx | xx | 0.xxx | xx | xx | 0.xxx |
| X | xx | xx | 0.xxx | xx | xx | 0.xxx |
| X | xx | xx | 0.xxx | xx | xx | 0.xxx |
| X | xx | xx | 0.xxx | xx | xx | 0.xxx |
| X | XX | xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | Xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | Xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | Xx | 0.xxx | XX | xx | 0.xxx |
| X | XX | Xx | 0.xxx | XX | XX | 0.xxx |
| X | XX | Xx | 0.xxx | xx | xx | 0.xxx |
| 25th percentile [1] | | xx.x | | | xx.x | |
| 50th percentile [1] | | xx.x | | | xx.x | |
| 75 <sup>th</sup> percentile [1] | | xx.x | | | xx.x | |
| p-value [2] | | x.xxxx | | | | |

 $n = number \ of \ participants \ with \ a \ confirmed \ undetectable \ assessment \ by \ the \ end \ of \ the \ period. \ N\# = number \ of \ participants \ at \ risk.$ 

- [1] Percentiles are obtained from the Kaplan-Meier estimates.
- [2] P-value obtained from a log-ank test compared RV299 and placebo.

Note: Time to First Confirmed Undetectable Assessment from Initial Administration of IMP = (Date of first confirmed negative test after peak qRT-PCR measurement - Date of first administration of IMP) + 1.

This table may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

This layout will be utilised for the following tables:

Table 14.2.2.3.1 Time to First Confirmed Undetectable Assessment of RSV Challenge Virus after Peak Measure by qRT-PCR from qRT-PCR following Initial Administration of IMP - ITT-I Population

Table 14.2.2.4.1 Time to Peak RSV Challenge Virus qRT-PCR following Initial Administration of IMP - ITT-I Population

Table 14.2.2.7.1 Time to First Confirmed Undetectable Assessment of RSV Challenge Virus after Peak Measure by Viral Culture starting from Initial Administration of IMP - ITT-I Population

Table 14.2.2.8.1 Time to First Confirmed Undetectable Assessment of RSV Challenge Virus by Viral Culture starting from Peak Measure - ITT-I Population

Where appropriate, these tables may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

Table 14.2.3.1.1

AUC of Total Symptom Score from 10-Item Diary Card from First Administration of IMP to Quarantine Discharge ITT-I Population

| | Treatmer | nt Group |
|----------------------------------------|----------------|--------------|
| AUC (hours*score) | RV299 | Placebo |
| | (N=xx) | (N=xx) |
| n | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| GM (GSD) | XX.X (XX.XX) | XX.X (XX.XX) |
| %CV | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, X.XX | XX.X, X.XX |
| Min, Max | XX, XX | XX, XX |
| Difference in LS means [1] | XX.XX | |
| 95% Confidence interval for difference | XX.XXX, XX.XXX | |
| P-value [1] | X.XXX | |

[1] Comparison of RV299 and placebo using an ANCOVA with treatment group as a fixed effect and baseline viral load as the covariate.

Note: Total symptom scores at the time of the first administration of IMP can be prior to or after dosing, depending on whether dosed in the morning or evening.

Note: GM is derived by antilog( mean( exp( TSS-AUC + 1 ) ) ) - 1.

This table may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

This layout will be utilised for the following tables:

Table 14.2.3.1.2 AUC of Total Symptom Score from 10-Item Diary Card from First Administration of IMP for 6.5 Days - ITT-I Population

Table 14.2.3.2.1 AUC of Total Symptom Score from 10-Item Diary Card from Day 2 to Day 12 - ITT-I Population

Table 14.2.3.2.1 AUC of Total Symptom Score Change from Baseline from 10-Item Diary Card from First Administration of IMP to Quarantine Discharge - ITT-I Population

Table 14.2.3.2.2 AUC of Total Symptom Score Change from Baseline from 10-Item Diary Card from First Administration of IMP for 6.5 Days - ITT-I Population

Table 14.2.3.2.3 AUC of Total Symptom Score Change from Baseline from 10-Item Diary Card from Day 2 to Day 12 - ITT-I Population

Table 14.2.3.4.1 Peak Total Symptom Score from 10-Item Diary Card from First Administration of IMP to Quarantine Discharge - ITT-I Population

Where appropriate, these tables will be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

Programming Note: It is highly likely that the parametric methods will fail to meet the required assumptions. Therefore, we will provide a Wilcoxon test (see Section 10.1.4). The alternative presentation for this is shown below and will require the following footnote update: [1] Comparison of RV299 and placebo using a Wilcoxon rank sum test.

Median difference in LS means [1] XX.XX P-value [1] X.XXX

Table 14.2.3.3.1
Total Symptom Score from 10-Item Diary Card by Assessment ITT-I Population

| | | Treatment Group | | | |
|---|---|---|---|---|---|
| | | | RV299<br>N=xx) | Plac<br>(N= | cebo<br>xx) |
| Days from IMP Administration<br>Assessment | Observed | | Change from Baseline | Observed | Change from<br>Baseline |
| ) Days | n | XX | | XX | |
| Assessment 1 | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | GM (GSD) | XX.X (XX.XX) | | XX.X (XX.XX) | |
| | %CV<br>Median | XX.XX<br>XX.X | | XX.XX<br>XX.X | |
| | Q1, Q3 | XX.X, X.XX | | XX.X, X.XX | |
| | Min, Max | XX, XX | | XX, XX | |
| O Days | n | XX | XX | XX | XX |
| Assessment 2 | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| | GM (GSD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX |
| | %CA | XX.XX | XX.XX | XX.XX | XX.XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Q1, Q3 | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX |

Note: Assessments are relative to first administration of IMP.

Note: Total symptom scores at the time of the first administration of IMP can be prior to or after dosing, depending on whether dosed in the morning or evening.

This table may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 respectively.

This layout will be utilised for the following tables:

Table 14.2.3.5.1 Peak Total Symptom Score from 10-Item Diary Card by Day - ITT-I Population

The table may be repeated on the ITT-A, ITT-B, ITT and PP Populations as .2, .3, .4 and .5 as appropriate.

Table 14.2.3.6.1

Peak Daily Symptom Score from 10-Item Diary Card
ITT-I Population

| | | | Treatment | Group | |
|---|---|---|---|---|---|
| | | | RV299<br>(N=xx) | | acebo<br>N=xx) |
| Days from IMP Administration | | Observed | Change from Baseline | Observed | Change from Baseline |
| 0 Days | n<br>Mean (SD)<br>GM (GSD)<br>%CV<br>Median<br>Q1, Q3<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X (XX.XX)<br>XX.XX<br>XX.X<br>XX.X, X.XX<br>XX, XX | | XX<br>XX.X (XX.XX)<br>XX.X (XX.XX)<br>XX.XX<br>XX.X<br>XX.X<br>XX.X, X.XX | |
| 1 Day | n<br>Mean (SD)<br>Median<br>GM (GSD)<br>%CV<br>Q1, Q3<br>Min, Max | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X (XX.XX)<br>XX.XX<br>XX.X, X.XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X (XX.XX)<br>XX.XX<br>XX.X, XXX<br>XX, XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X (XX.XX)<br>XX.XX<br>XX.X, X.XX | XX<br>XX.X (XX.XX)<br>XX.X<br>XX.X (XX.XX)<br>XX.XX<br>XX.X, X.XX<br>XX, XX |

Note: Days are relative to first administration of IMP.

Note: Total symptom scores on the day of the first administration of IMP can be prior to or after dosing, depending on whether dosed in the morning or evening.

Table 14.2.3.7.1

Time to Symptom Resolution by 10-Item Diary Card from Initial Administration of IMP to 24-Hours Symptom Free ITT-I Population

| | Treatme | Treatment Group |
|-------------|--------------|-----------------|
| | RV299 | Placebo |
| Time (days) | (N=xx) | (N=xx) |
| n | XX | XX |
| Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) |
| GM (GSD) | XX.X (XX.XX) | XX.X (XX.XX) |
| %CV | XX.XX | XX.XX |
| Median | XX.X | XX.X |
| Q1, Q3 | XX.X, X.XX | XX.X, X.XX |
| Min, Max | XX, XX | XX, XX |

Note: Time to Symptom Resolution from Initial Administration of IMP = (Date and time of symptom resolution - Date of and time of assessment at time of IMP administration) + 1.

This layout will be utilised for the following tables:

Table 14.2.3.8.1 Time to Symptom Resolution by 10-Item Diary Card from Peak Total Symptom Score to 24-Hours Symptom Free - ITT-I Population Table 14.2.3.9.1 Time to Peak Symptom Score by 10-Item Diary Card from Initial Administration of IMP - ITT-I Population

The layout will be repeated for the following tables, without the GM (GSD) row:

Table 14.2.4.1.1 Total Weight of Mucus Produced from Initial Administration of IMP to Quarantine Discharge - ITT-I Population

Table 14.2.4.2.1 Total Number of Tissues Used from Initial Administration of IMP to Quarantine Discharge by Assessment - ITT-I Population



Table 14.3.1.67

Overall Summary of Treatment Emergent Adverse Events
Safety Population

| | Treatment Group | | | | | |
|---|---|---|---|---|---|---|
| | | RV299<br>N=xx) | | cebo<br>xxx) | | rerall<br>N=xx) |
| | n | (%) | n | (%) | n | (%) |
| umber of Events | XX | | XX | | XX | |
| umber of Participants with any Adverse Event | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| umber of Participants with any Serious Adverse Event | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| umber of Participants with any Related Adverse Event | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| umber of Participants with any Adverse Event Leading<br>o Withdrawal from the Study | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |
| umber of Participants with any Adverse Event Leading o Discontinuation of IMP | XX | (XX.X) | XX | (XX.X) | XX | (XX.X) |

Note: Treatment emergent events are those events with an onset on or after the start of IMP dosing.

Note: If a participant experiences more than one event, then the event with the worst severity or strongest relationship is included in the relevant level of summarisation.

Note: Related = 'Unlikely', 'Possibly', 'Probably', 'Definitely' or 'Not assessed'.

Note: Adverse Event Leading to Discontinuation from the Study = Participant withdrew from the study due to an adverse event.

Note: Adverse Event Leading to Discontinuation of Dosing = Action taken of 'Trial/Study drug permanently discontinued'.

Table 14.3.1.68

Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Population

| | Treatment Group | | | |
|---|---|---|---|---|
| | 1 | RV299 | Pla | acebo |
| System Organ Class/ | ( | (N=xxx) | | |
| Preferred Term [1] | n | (%) | n | (%) |
| Number of Events | XX | | XX | |
| Number of Subjects with any adverse event | XX | (XX.X) | XX | (XX.X) |
| System Organ Class 1 | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 2 | XX | (XX.X) | XX | (XX.X) |
| System Organ Class 2 | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 2 | XX | (XX.X) | XX | (XX.X) |

Note: Treatment emergent events are those events with an onset on or after the first administration of IMP.

Note: Table shows distinct number of participants with events for each system organ class/preferred term.

<sup>[1]</sup> MedDRA Version 25.0.

 ${\small \mbox{Table 14.3.1.3}}$  Treatment Emergent Adverse Events by System Organ Class, Preferred Term and Severity Safety Population

| | | Treatmen | nt Group | |
|----------------------|----|----------|----------|--------|
| | ] | RV299 | Pla | cebo |
| System Organ Class/ | ( | N=xx) | (N=xxx) | |
| Preferred Term [1] | n | (%) | n | (%) |
| System Organ Class 1 | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 2 | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) |
| System Organ Class 2 | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Mild | XX | (XX.X) | XX | (XX.X) |
| Moderate | XX | (XX.X) | XX | (XX.X) |
| Severe | XX | (XX.X) | XX | (XX.X) |

#### [1] MedDRA Version 25.0.

Note: Treatment emergent events are those events with an onset on or after the first administration of IMP.

Note: This table shows distinct number of participants with events for each system organ class/preferred term/severity. If a participant experienced a specific event more than once then the event with the worst severity is summarised.

Table 14.3.1.4

Treatment Emergent Adverse Events Related to RV299 by System Organ Class and Preferred Term
Safety Population

| | Safety Population | Treatme | nt Group | |
|---|---|---|---|---|
| System Organ Class/ | ī | RV299 | - | cebo |
| Preferred Term [1]/ | | (N=xx) | | (N=xxx) |
| Relationship | 'n | (%) | n (N- | (%) |
| noracronomp | ** | (0) | | (0) |
| System Organ Class 1 | XX | (XX.X) | XX | (XX.X) |
| Not Assessed | XX | (XX.X) | XX | (XX.X) |
| Unlikely Related | XX | (XX.X) | XX | (XX.X) |
| Possibly Related | XX | (XX.X) | XX | (XX.X) |
| Probably Related | XX | (XX.X) | XX | (XX.X) |
| Definitely Related | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Not Assessed | XX | (XX.X) | XX | (XX.X) |
| Unlikely Related | XX | (XX.X) | XX | (XX.X) |
| Possibly Related | XX | (XX.X) | XX | (XX.X) |
| Probably Related | XX | (XX.X) | XX | (XX.X) |
| Definitely Related | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 2 | XX | (XX.X) | XX | (XX.X) |
| Not Assessed | XX | (XX.X) | XX | (XX.X) |
| Unlikely Related | XX | (XX.X) | XX | (XX.X) |
| Possibly Related | XX | (XX.X) | XX | (XX.X) |
| Probably Related | XX | (XX.X) | XX | (XX.X) |
| Definitely Related | XX | (XX.X) | XX | (XX.X) |
| System Organ Class 2 | XX | (XX.X) | XX | (XX.X) |
| Not Assessed | XX | (XX.X) | XX | (XX.X) |
| Unlikely Related | XX | (XX.X) | XX | (XX.X) |
| Possibly Related | XX | (XX.X) | XX | (XX.X) |
| Probably Related | XX | (XX.X) | XX | (XX.X) |
| Definitely Related | XX | (XX.X) | XX | (XX.X) |
| Preferred Term 1 | XX | (XX.X) | XX | (XX.X) |
| Not Assessed | XX | (XX.X) | XX | (XX.X) |
| Unlikely Related | XX | (XX.X) | XX | (XX.X) |
| Possibly Related | XX | (XX.X) | XX | (XX.X) |
| Probably Related | XX | (XX.X) | XX | (XX.X) |
| Definitely Related | XX | (XX.X) | XX | (XX.X) |

Note: Treatment emergent events are those events with an onset on or after the first administration of IMP.

Note: This table shows distinct number of participants with events for each system organ class/preferred term/relationship. If a participant experiences a specific event more than once then the event with the greatest relationship is summarised.

Note: Only the subset of AEs that are judged to be related to IMP have been considered (i.e. relationship = Possibly Related/Probably Related/Definitely Related/Not Assessed) in the table.

Note: Percentages are based on the safety population.

This layout will be utilised for the following table:

Table 14.3.1.5 Adverse Events Related to Challenge Agent by System Organ Class and Preferred Term - Safety Population With the following footnote:

Note: Only the subset of AEs that are judged to be related to challenge agent have been considered (i.e. relationship = Possibly Related/Probably Related/Definitely Related/Not Assessed) in the table.

<sup>[1]</sup> MedDRA Version 25.0.

Table 14.3.2 Haematology Parameters: Summary Safety Population

| | | Treatment Group | | | | |
|---|---|---|---|---|---|---|
| | | RV299<br>(N=xx) | | Placebo<br>(N=xx) | | |
| | | | | | | Parameter (units) |
| Baseline | n | XX | | XX | | |
| | Mean (SD) | XX.X (XX.XX) | | XX.X (XX.XX) | | |
| | %CV | xx.xx | | XX.XX | | |
| | Median | XX.X | | XX.X | | |
| | Q1, Q3 | XX.X, X.XX | | XX.X, X.XX | | |
| | Min, Max | XX, XX | | XX, XX | | |
| Day 7 | n | XX | XX | XX | XX | |
| - | Mean (SD) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | XX.X (XX.XX) | |
| | %CV | XX.XX | XX.XX | XX.XX | XX.XX | |
| | Median | XX.X | XX.X | XX.X | XX.X | |
| | Q1, Q3 | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX | XX.X, X.XX | |
| | Min, Max | XX, XX | XX, XX | XX, XX | XX, XX | |

This layout will be utilised for the following tables:

| Table 14.3.3 | Biochemistry Parameters: Summary - Safety Population |
|---|---|
| Table 14.3.4 | Coagulation Parameters: Summary - Safety Population |
| Table 14.3.5 | Cardiac Enzyme Parameters: Summary - Safety Population |
| Table 14.3.6 | Urinalysis Parameters: Summary - Safety Population |
| Table 14.3.7 | Vital Signs Parameters: Summary - Safety Population |
| Table 14.3.8 | Spirometry Parameters: Summary - Safety Population |
| Table 14.3.9 | 12-Lead Electrocardiogram Parameters: Summary - Safety Population |

Listing 16.2.1.1 Participant Disposition

| Treatment<br>Group | Participant<br>Number /<br>Randomisation<br>Number | Date/Time of Informed Consent: V2 / V3 / V5.1 / V8 / Genetic testing V1 / Genetic testing V2 | Date/Time of: Quarantine Admission / Randomisation / Challenge Agent Administration / First IMP Administration / Quarantine Discharge | Eligible for randomisation? [1] /<br>Completed IMP? /<br>Completed Study? [2] | Reason not randomized /<br>Reason for discontinuation of IMP /<br>Reason for withdrawal |
|---|---|---|---|---|---|
| xxxxxx | xxxxxx /<br>xxxxxx | ddmmmyyyy hh:mm / NA / ddmmmyyyy hh:mm / ddmmmyyyy hh:mm / NA / ddmmmyyyy hh:mm | ddmmmyyyy hh:mm / ddmmmyyyy hh:mm / ddmmmyyyy hh:mm / ddmmmyyyy hh:mm / ddmmmyyyy hh:mm | Yes or No /<br>Yes or No /<br>Yes or No | XXXXXXXXXXXXXXXXX /<br>XXXXXXXXXXXXXXXXXX /<br>XXXXXXXX |

NA = Not applicable.
[1] Eligible for randomisation based on criteria at Admission (Day -2/-1).
[2] Completed Study = Participating in the study up to and including Day 28 (Follow-up).
Listing 16.2.1.2 Failed Inclusion and Exclusion Criteria

| Treatment Group | Participant | Reason for Exclusion |
|-----------------|-------------|----------------------|
| xxxxxxx | xxxxxx | xxxxxxxxxxxxxxxx |

Programming note: Listing not required if no participants fail the criteria.

Listing 16.2.74 Protocol Deviations

| Treatment | Participant | Deviations | Date Occurred | Deviation | Other, | Deviation | Serious |
|---|---|---|---|---|---|---|---|
| Group | | Reported | (Study Day) | Category [a] | Specify | Description | Breach? |
| xxxxxx | xxxxxx | Yes/No | ddmmmyyyy (xx) | n | xxxx | xxxxxxxxx | Yes / No |

[a] - Deviation categories: Informed Consent procedure [1] / Subject error [2] / Inclusion/exclusion criteria [3] / Investigational product [4] / Visit window [5] / Concomitant medication/therapy [6] / Study procedure/assessment window [7] / SAE reporting [8] / Study procedure/assessment performance [9] / Randomisation [10] / Missing assessment/sample [11] / Other [12]

# Listing 16.2.75 Participant Populations

| Treatment Group | Participant | ITT<br>Population [1] | ITT-I<br>Population [2] | ITT-A<br>Population [3] | ITT-B<br>Population [4] | PP Population<br>[5] | Safety<br>Population [6] | PK Population<br>[7] |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | Yes / No | Yes / No | Yes / No | Yes / No | Yes / No | Yes / No | Yes / No |

[1] Intent to Treat (ITT) Population = All randomised participants receiving challenge virus and at least one dose IMP

[2] Intent to Treat Infected (ITT-I) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection. A laboratory-confirmed RSV infection is defined as the presence of viral shedding, measured in nasal wash where one or both of the following definitions must be met: At least 2 positive detections by viral load qRT-PCR assay specific for the challenge virus, reported on 2 or more consecutive days; One positive detection by viral load qRT-PCR assay, specific for the challenge virus, in which an aliquot of the same sample has also tested positive in a cell-based assay appropriate for detecting the challenge virus.

[3] Intent to Treat Infected Pre-dose (ITT-A) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection, using only assessments prior to taking IMP.

[4] Intent to Treat Infected Post-dose (ITT-B) Population = All randomised participants receiving challenge virus and at least 1 dose of IMP, and meeting the criterion for laboratory confirmed RSV infection, using only assessments after IMP.

[5] Per Protocol (PP) Population = All ITT-I population participants who have no major protocol deviations, and who complete the quarantine period up to the final day of quarantine (Study Day 12) and receive all 10 doses of IMP.

[6] Safety Population = All randomised participants receiving challenge virus and at least one dose of IMP.

[7] The PK Population = All ITT participants with at least one post-dose PK result.

Listing 16.2.4.76 Demographics

| Treatment<br>Group | Participant | Age at Time of screening (years) | Sex | Race / Ethnicity | Visit | Date / Time | Height<br>(cm) | Weight<br>(kg) | BMI<br>(kg/m^2) | Comments |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | хх | Male /<br>Female | xxxxxx / xxxxxx | Screening | ddmmmyyyy / hh:mm | xxx | xx.xx | xx | xxxxxx |

NA = Not Applicable.

Note: Results for height, weight and BMI are shown for all visits at which they were recorded.

Programming note: For height, weight, and BMI if recording is repeated, then all sets of results should be shown.

#### Listing 16.2.4.77 Reproductive Status and Contraceptive Use

| Treatment<br>Group | Participant | Sex | Breast Feeding/<br>Pregnant Recently<br>/<br>Planning<br>Pregnancy | Child-bearing potential? | Agree to not donate sperm | (Hetero)<br>Sexually<br>active? | Agree to contraception | Contraception methods [1] |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Male<br>Female | NA<br>Yes / No | NA<br>Yes /<br>No; menopausal /<br>No; incapable | Yes / No<br>NA | Yes / No<br>Yes / No | Yes / No<br>Yes / No | 1 3 |

- [1] 1 Male sterilisation where vasectomised male is the sole partner for that woman.

  - 2 Oral, injected or implanted hormonal methods of contraception (minimum 2 weeks prior to admission).

    3 An intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) or bilateral tubal ligation.
  - 4 Male condom with spermicide and female partner using a highly effective method of contraception (e.g. IUD, IUS, bilateral ligation).

Listing 16.2.4.78 Smoking History

| Treatment<br>Group | Participant | Smoking History | Start Date | Stop Date | Date Last<br>Smoked | Category | Amount | Years | Comments |
|---|---|---|---|---|---|---|---|---|---|
| XXXXXXX | XXXXXX | XXXXXXXXX | ddmmyyyy | ddmmyyyy | ddmmyyyy | Number of cigarettes smoked per day | XX | XX | XXXXXXXXXX |
| | | | | | | Number of cigars smoked per day | XX | XX | XXXXXXXXXX |
| | | | | | | Tobacco smoked per week (grams) | xx | xx | xxxxxxxxxx |
| | | | | | | Pack years | xx | xx | xxxxxxxxxx |

<sup>\*</sup> Date estimated.

Note: Comments are collected for the combined smoking, alcohol and drugs of abuse module and hence may relate to any of these parameters.

Listing 16.2.4.79
Alcohol Use

| Treatment<br>Group | Participant | Alcohol Use History | Weekly alcohol intake (units) | Willing to refrain from alcohol intake | Comments |
|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Never / Current User / | xx | Yes / No | xxxxxxxxx |

Note: Comments are collected for the combined smoking, alcohol and drugs of abuse module and hence may relate to any of these parameters.

#### Listing 16.2.4.80 Recreational Drugs of Misuse

| Treatment<br>Group | Participant | Current or recent user of recreational drugs? | Start Date | Stop Date | Recreational drug(s) used | Volume | Route | Comments |
|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Yes / No | ddmmmyyyy* | ddmmmyyyy / hh:mm | XXXX | XXXX | XXXX | XXXX |

NA = Not Applicable. \* = Date estimated.

Listing 16.2.4.81 Medical History

| Treatment<br>Group | Participant | MedDRA SOC /<br>Preferred Term [1] /<br>Medical Condition | Start Date<br>/ End Date | Line No. | Frequency | Ongoing | Concomitant medication taken for this condition? |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Xxxxxxxx<br>Xxxxxxxx<br>Xxxxxxxxx | ddmmmyyyy /<br>ddmmmyyyy | xxxx | Single Episode /<br>Intermittent /<br>Continuous /<br>Other | Yes / No | Yes / No |

<sup>\*</sup> Date estimated.

<sup>[1]</sup> MedDRA Version 25.0. The modified term is the term that was used for MedDRA coding of the event when the event required multiple codes.

# Listing 16.2.4.82 Prior and Concomitant Medications

| Treatment<br>Group | Participant | Drug Class (L2)/<br>WHO Drug Name/<br>Medication (verbatim)[1] | Start Date<br>/ Time | Stop Date<br>/ Time | Ongoing | Indication / AE/ Medical History Line | Dose /<br>Dose<br>units | Frequency [2] | Route<br>[3] | PI / P /<br>C [4] |
|---|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | Xxxxxxxx<br>Xxxxxxxx | ddmmmyyyy /<br>hh:mm | ddmmmyyyy /<br>hh:mm | Yes / No | Xxxxxxxxx /<br>Xxxxxxxxx / | XX xx | XXX | XXX | PI |
| | | Xxxxxxxx | hh:mm | hh:mm | | Xxxxxxxxx /<br>Xxxxxxxxx | | | | |

<sup>\* =</sup> Date/time estimated.

<sup>[1]</sup> WHO Drug Global Version 2022:1, March 1, 2022.

<sup>[2]</sup> QD = Once a day, BD = Twice a day, PRN = As needed, TDS = Three times a day, QDS = Four times a day.

<sup>[3]</sup> PO = oral, TOP = topical, PRN = Take as needed.

<sup>[4]</sup> PI = Prior to Inoculation, P = Prior to IMP treatment and after inoculation, C = Concomitant with IMP treatment.

Note: If the medication stop date is before the date of inoculation the medication will be assigned as prior to inoculation. If the medication stop date is before the date of IMP treatment but after the date of inoculation, the medication will be assigned as being prior to IMP treatment. In all other cases, the medication is assigned as concomitant with IMP treatment.

#### Listing 16.2.5.83 Challenge Virus Inoculation Administration

| Treatment<br>Group | Participant | Administration<br>Date / Time | Administered intranasally? | Administered to both nostrils? | Administered successfully? | Change in health in 30 minutes post administration? | Comments |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | ddmmmyyyy / hh:mm | Yes / No | Yes / No | Yes / No | Yes / No | XXXXXXX |

#### Listing 16.2.5.84 Viral Shedding Results

| Treatment<br>Group | Participant | Study day and nasal wash time-point | qicPCR result | Comments |
|---|---|---|---|---|
| xxxxxx | xxxxx | Day X AM/PM<br>Day X AM/PM | Positive/Negative/Invalid/NA<br>Positive/Negative/Invalid/NA | XXXXXXXX |
| | | <br>Subject to be dosed Day 5 PM | NA | XXXXXXXX |

Listing 16.2.5.3 IMP Administration

| Treatment<br>Group | Participant | Dose<br>Number | | | Was dose fully administered? | Comments |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XX | Yes / No | ddmmmyyyy / hh:mm | Yes / No | XXXXXXXX |

Listing 16.2.6.1.1
Viral Load by Nasal Samples qRT-PCR Results

| Treatment<br>Group | Participant | Sample Collection<br>Date / Time<br>(Study Day) | Assessment | Virus Titre<br>(Log10 Copies/mL) | Did<br>Participant<br>Bleed? | Comments |
|---|---|---|---|---|---|---|
| xxxxxxx | xxxxx | ddmmyyyy / hh:mm | 1 / 2 | Xxxxx | Yes / No | xxxxxxxxxx |

Programming Note: The Limit of Detection and Lower limit of Quantification will be shown in the footnote.

Listing 16.2.6.1.2
Viral Load by Nasal Samples qRT-PCR Derivations

| Treatment<br>Group | Participant | IMP administration<br>to planned discharge<br>(hours*Log10<br>Copies/mL) | AUC<br>IMP administration<br>for 6.5 days<br>(hours*Log10<br>Copies/mL) | Day 2 to Day 12<br>(hours*Log10<br>Copies/mL) | IMP administration<br>to planned discharge<br>(hours*Copies/mL) | Peak Viral Load<br>(from IMP<br>administration to<br>Day 12)<br>(Log10 Copies/mL) | Time from IMP<br>administration<br>to negative<br>test after Peak<br>measure (days) | Time from Peak measure after IMP administration to negative test after peak measure (days) | Time to<br>Peak<br>Measure<br>(days) |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxx | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX | XX | XX |

Note: For the calculation of AUCs, values that are 'Not Detected', 'Detected' or are at or below the limit of quantification have been re-assigned to 0.

<sup>\* =</sup> Censored value.

Listing 16.2.6.2.1
Viral Load by Nasal Samples Viral Culture Results

| Treatment<br>Group | Participant | Sample<br>Type | Sample Collection<br>Date / Time<br>(Study Day) | Assessment | Virus Titre<br>(Log10 Copies/mL) | Comments |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | Xxxxxxxxx | ddmmyyyy / hh:mm (xx) | 1 / 2 | xxxx | xxxxxxxxxxxxxxxx |

Programming Note: The Limit of Detection and Lower limit of Quantification will be shown in the footnote.

Listing 16.2.6.2.2

| | | | Vira | al Load by Nasal Sar | mples Viral Culture I | erivations | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | AUC | | | Peak Viral Load | | Time from Peak | |
| | | IMP administration | IMP administration | | IMP | (from IMP | Time from IMP | measure after IMP | Time to |
| Treatment | | to planned discharge (hours*Log10 | for 6.5 days<br>(hours*Log10 | Day 2 to Day 12<br>(hours*Log10 | administration to planned discharge | administration to Day 12) | administration to<br>negative test after | administration to<br>negative test after | Peak<br>Measure |
| Group | Participant | Copies/mL) | Copies/mL) | Copies/mL) | (hours*Copies/mL) | (Log10 Copies/mL) | Peak measure (days) | peak measure (days) | (days) |
| XXXXXXX | XXXXXX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX | XX | XX |

Note: For the calculation of AUCs, values that are 'Not Detected', 'Detected' or are at or below the limit of quantification have been re-assigned to 0.

<sup>\* =</sup> Censored value.

#### Listing 16.2.6.3.1 Symptom Scores from Symptom Diary Card

| Treatment<br>Group | Participant | Diary Card Completion Date / Time (Study Day) | Days from IMP<br>Administration | Assessment | LRT<br>Grades<br>[1] | URT<br>Grades<br>[2] | S Grades | 10-item<br>Score [ | Symptom | 13-item<br>Score | Symptom |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Total | CFB | Total | CFB |
| xxxxxx | xxxxx | ddmmyyyy /<br>hh:mm | XX | 1 / 2 / 3 | X/X/X/X | X/X/X/X/<br>X | X/X/X/X | xx | xx | xx | xx |

LRT = Lower respiratory tract. URT = Upper respiratory tract. S = Systemic. CFB = Change from Baseline.

<sup>[1]</sup> Cough/Shortness of Breath/Chest Tightness/Wheeze

<sup>[1]</sup> Cough/Shortness of Breath/Chest Tightness/Mneeze
[2] Runny Nose/Stuffy Nose/Sneezing/Sore Throat/Earache
[3] Headache/Malaise/Muscle Joint, Ache/Chilliness, Feverishness
[4] Includes Cough/Shortness of Breath/Runny Nose/Stuffy Nose/Sneezing/Sore Throat/Earache Headache/Malaise/Muscle Joint, Ache. Note: A total symptom score requires at least one symptom to be scored.

#### Listing 16.2.6.3.2 Visual Analogue Scale from Symptom Diary Card

| Treatment<br>Group | Participant | Diary Card Completion<br>Date / Time<br>(Study Day) | Days from IMP<br>Administration | Assessment | LRT<br>Grades<br>(mm)[1] | URT<br>Grades<br>(mm)[2] | S Grades<br>(mm) [3] |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | ddmmyyyy / hh:mm | XX | 1 / 2 / 3 | XX/XX/XX<br>/XX | XX/XX/XX<br>/XX/XX | XX/XX/XX/<br>XX |

LRT = Lower respiratory tract. URT = Upper respiratory tract. S = Systemic. [1] Cough/Shortness of Breath/Chest Tightness/Wheeze

<sup>[2]</sup> Runny Nose/Stuffy Nose/Sneezing/Sore Throat/Earache
[3] Headache/Malaise/Muscle Joint, Ache/Chilliness, Feverishness

# Listing 16.2.6.3.3 Total Symptom Score: AUC Derivations

| | | Total Symptom Score AUC [1] | | | Total Symptom Sco. | re Change from Base | eline AUC | Total Symptom Score AUC [2] | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Participant | IMP<br>administration to<br>planned discharge | IMP<br>administration<br>for 6.5 days | Day 2 to<br>Day 12 | IMP<br>administration to<br>planned discharge | IMP<br>administration<br>for 6.5 days | Day 2 to<br>Day 12 | IMP<br>administration to<br>planned discharge | IMP<br>administration<br>for 6.5 days | Day 2 to<br>Day 12 |
| xxxxxxx | xxxxxx | XX | XX | XX | XX | XX | XX | XX | XX | XX |

<sup>[1]</sup> Derivations made using 10-items of the 13-item symptom diary card.

<sup>[2]</sup> Derivations made using all 13-items of the symptom diary card.

# Listing 16.2.6.3.4 Total Symptom Score: Other Derivations

| | | Days from | Sum Total<br>Symptom Score<br>(from IMP | Peak Total<br>Symptom Score<br>(from IMP | Peak Daily Total<br>Symptom Score<br>(from IMP | Time to Symptom<br>Resolution from | Time to Symptom<br>Resolution from<br>Peak Symptom | Time to Peak<br>Total Symptom |
|---|---|---|---|---|---|---|---|---|
| Treatment<br>Group | Participant | IMP<br>Administra<br>tion | administration to planned discharge) | administration to planned discharge) | administration to planned discharge) | IMP<br>administration<br>(days) | after IMP<br>administration<br>(days) | Score from IMP administration (days) |
| ×××××× | ×××××× | XX | XX | XX | XX | XX | XX | XX |

Note: Derivations made for 10-items of the 13-item diary card.

Programming Note: Place the endpoints that are not by study day onto the first row for each participant.

# Listing 16.2.6.4.1 Mucus Weight and Tissue Bag Distribution

| Treatment<br>Group | Participant | Study Day | Date<br>Collected | Tissue Bag Distribution Time Collected/Dispensed | Tissues<br>Taken | Total Tissues<br>Taken | Mucus Weight (g) | Total Mucus Weight (g) | Comments |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | xx | ddmmyyyy | hh:mm | xxxx | xxxx | xxxx | xxxx | |

Programming note: The Total Mucus Weight and Total Tissues Taken will be listed against the Day 12 observation.

Listing 16.2.6.5.1
Nasopharyngeal Swab: Respiratory Virus Screen/Rapid Viral Antigen Test

| Treatment<br>Group | Participant | Sample Collection<br>Date / Time<br>(Study Day) | Result | Comments |
|---|---|---|---|---|
| xxxxxx | xxxxxx | ddmmyyyy / hh:mm (xx) | Positive / Negative | xxxxxxx |

Listing 16.2.6.6 Plasma PK Parameters

| Treatment<br>Group | Participant | Day | PK Parameter | Units | RV299 | Comments |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | XXX | XXX | XXX | XXX | xxxxxxx |

Listing 16.2.7 Adverse Events

| Treatment<br>Group /<br>Participant<br>/AE Number | MedDRA SOC / Preferred Term [1] / Adverse event (verbatim) | Start Date Time<br>(study day) /<br>Stop Date Time<br>(Study day) | TE [2] /<br>CE [3] /<br>Severity /<br>Frequency [4] | SAE /<br>Serious<br>Criteria [5] | Outcome [6] /<br>Action Taken IMP [7] /<br>Action Taken [8] / | Related to [9] IMP / Challenge Agent / Concomitant medication / Procedure / Other | Comments |
|---|---|---|---|---|---|---|---|
| xxxxxxx /<br>xxxx / xx | xxxxxxxx/<br>xxxxxx/<br>xxxxxx | ddmmmyyyy hh:mm (xx) / ddmmmyyyy hh:mm (xx) | Yes or No / Yes or No / Mild, Moderate, Severe, Life- Threatening / | Yes or Blank / xx | x /<br>x /<br>x | x / x / x / x / x | XXXXXXXXXXX |

TE = Treatment Emergent. SAE - Serious Adverse Event.

- [1] MedDRA Version 24.0.
- [2] An AE occurring on or after the first administration of IMP.
- [3] An AE occurring on or after the challenge agent inoculation.
- [4] Freq = Frequency. For frequency categories, C = Continuous, I = Intermittent, S = Single Episode.
- [5] Serious Criteria: 1 = Death; 2 = Life-threatening; 3 = Hospitalization; 4 = Persistent or significant disability/incapacity; 5 = Congenital anomaly/birth defect; 6 = Other.
- [6] Outcome: 1 = Resolved; 2 = Resolved with Sequelae; 3 = Ongoing; 4 = Fatal; 5 = Unknown.
- [7] Action Taken IMP: 1 = IMP dosage not changed; 2 = IMP dosage adjusted; 3 = IMP administration temporarily interrupted; 4 = IMP administration discontinued.
- [8] Action Taken: 1 = None; 2 = Non-drug therapy given; 3 = Concomitant medication taken; 4 = Participant withdrawn; 5 = Participant hospitalized; 6 = Other; 7 = Not applicable.
- [9] Related: 1 = Not Related; 2 = Unlikely Related; 3 = Possibly Related; 4 = Probably Related; 5 = Definitely Related.

#### Listing 16.2.8.98 Blood Sample Collection

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Sample Type(s) [1] | Clinically<br>Significant<br>Result? | Adverse Event<br>associated with<br>Procedure? | Comments |
|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | | ddmmyyyy / hh:mm (xx) | x x x x x x | Yes / No | Yes / No | xxxxxxxxxxxx |

<sup>\*</sup> see Time and Events Schedule.

<sup>[1] 1 =</sup> Biochemistry, 2 = Cardiac enzymes, 3 = Haematology, 4 = Coagulation, 5 = Thyroid function test,

<sup>6 =</sup> Hepatitis B, & C, HIV serology, 7 = Serum pregnancy test, 8 = Serum follicle-stimulating hormone, 9 = Serum markers humoral immunity, 10 = Paxgene.

Listing 16.2.8.99
Haematology

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Parameter | Result | Change from<br>Baseline | Units | Lower<br>Limit | Upper<br>Limit | Flag | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | ddmmyyyy | | | | | | | | |
| | | | hh:mm | | | | | | | | |
| XXXXXXX | XXXXXX | XXXX | (xx) | Basophils (%) | X.XX | X.XX | % | X.XX | x.xx | L / H | xxxxxxxxxxxxxxxxxx |
| | | | | Basophils (abs) | x.xx | X.XX | X10^9/L | x.xx | x.xx | | |
| | | | | Eosinophils (%) | x.xx | X.XX | % | x.xx | x.xx | | |
| | | | | Eosinophils (abs) | x.xx | X.XX | X10^9/L | x.xx | x.xx | | |
| | | | | Haematocrit | x.xx | X.XX | ક | XX | XX | | |
| | | | | Haemoglobin | XXX | XXX | g/L | XXX | XXX | | |
| | | | | Lymphocytes (%) | x.xx | x.xx | % | x.xx | x.xx | | |
| | | | | Lymphocytes (abs) | x.xx | x.xx | X10^9/L | x.xx | x.xx | | |
| | | | | MCH | x.xx | x.xx | pg | xx.x | xx.x | | |
| | | | | MCHC | xxx | xxx | g/L | xxx | xxx | | |
| | | | | MCV | x.xx | x.xx | fL | xx.x | xx.x | | |
| | | | | Monocytes (%) | x.xx | x.xx | 8 | xx.x | xx.x | | |
| | | | | Monocytes (abs) | x.xx | x.xx | X10^9/L | xx.x | xx.x | | |
| | | | | Neutrophils (%) | x.xx | x.xx | % | xx.x | xx.x | | |
| | | | | Neutrophils (abs) | x.xx | x.xx | X10^9/L | xx.x | xx.x | | |
| | | | | Platelets | xxx | XXX | X10^9/L | xx.x | xx.x | | |
| | | | | RBC Count | x.xx | x.xx | X10^12/L | x.xx | x.xx | | |
| | | | | Reticulocytes (%) | x.xx | x.xx | % | x.xx | x.xx | | |
| | | | | Reticulocytes (abs) | xx.x | XX.X | X10^9/L | xx.x | xxx.x | | |
| | | | | WBC Count | x.xx | x.xx | X10^9/L | x.x | xx.x | | |

L = below lower limit, H = above upper limit.

This layout will be utilised for the following listings:

Listing 16.2.8.3 Coagulation

Listing 16.2.8.4 Biochemistry

Listing 16.2.8.5 Cardiac Enzymes

Listing 16.2.8.6 Thyroid Function Tests

Listing 16.2.8.100 Other Laboratory Tests: TDL

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Test | Result |
|---|---|---|---|---|---|
| | | | ddmmmyyyy / | | |
| | | | hh:mm | HIV 1 and HIV | 2 |
| xxxxxxx | xxxxxx | xxxx | (xx) | antibodies | Positive / Negative |
| | | | (/ | Hepatitis A | |
| | | | | Hepatitis B | |
| | | | | Hepatitis C | Positive / Negative |
| | | | | FSH | xx.x |
| | | | | Beta HCG | |
| | | | | (IU/L) | Positive / Negative |
| | | | | Immunoglobulin | |
| | | | | A antibodies | xx.x |
| | | | | HbA1C (%) | xx.x |
| | | | | HbA1C | |
| | | | | (mmol/mol) | xx.x |

L = Low, H = High, ND = Not Done.

Programming Note: Normal Ranges to be displayed in footnote, if available.

#### Listing 16.2.8.101 Other Laboratory Tests: Urine Pregnancy

| Treatment<br>Group | Participant | Visit | Test Date / Time<br>(Study Day) | Participant<br>has data | Result | Comments |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxx | xxxx | ddmmyyyy /<br>hh:mm<br>(xx) | Yes / No / NA - Male | Positive / Negative | xxxxxxxxxxxxxxx |

Listing 16.2.8.9.2 Other Laboratory Tests: Drugs of Abuse Screen

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Test<br>Performed<br>Time | Drug | Result | Comments |
|---|---|---|---|---|---|---|---|
| xxxxxxx | xxxxxx | xxxx | ddmmmyyyy | hh:mm | | Positive / | |
| ^^^^ | ΑΛΛΛΛΛ | AAAA | hh:mm | 1111.11411 | Cocaine | Negative / | |
| | | | (xx) | | COCATHE | Not done | |
| | | | (AA) | | | Positive / | |
| | | | | | Cannabinoids | Negative / | |
| | | | | | Calillabilioids | Not done | |
| | | | | | | Positive / | |
| | | | | | Methadone | Negative / | |
| | | | | | Mechadone | Not done | |
| | | | | | | Positive / | |
| | | | | | Ecstasy | Negative / | |
| | | | | | Ecocasy | Not done | |
| | | | | | | Positive / | |
| | | | | | Opiates | Negative / | |
| | | | | | Opiaces | Not done | |
| | | | | | | Positive / | |
| | | | | | Benzodiazepines | Negative / | |
| | | | | | Denzourazeprnes | Not done | |
| | | | | | | Positive / | |
| | | | | | Barbituates | Negative / | |
| | | | | | | Not done | |
| | | | | | | Positive / | |
| | | | | | Amphetamine | Negative / | |
| | | | | | 1 | Not done | |
| | | | | | | Positive / | |
| | | | | | Methamphetamine | Negative / | |
| | | | | | 1 | Not done | |
| | | | | | | Positive / | |
| | | | | | Tricyclic | Negative / | |
| | | | | | _ | Not done | |

# Listing 16.2.8.9. Other Laboratory Tests: Urine Cotinine

| Treatment<br>Group | Participant | Visit | Test Performed<br>Date / Time<br>(Study Day) | Result | Comments |
|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxx | ddmmyyyy / hh:mm (xx) | Positive / Negative | xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

# Listing 16.2.8.9. Other Laboratory Tests: Alcohol Breath Test

| Treatment | | _ | Test Date / Time | | |
|---|---|---|---|---|---|
| Group | Participant | Visit | (Study Day) | Result | Comments |
| xxxxxx | xxxxx | xxxx | ddmmyyyy / hh:mm | Positive / Negative | ****** |

Listing 16.2.9. Urinalysis

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Test Performed Time | Parameter | Result [1] |
|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxx | ddmmyyyy /<br>hh:mm<br>(xx) | hh:mm | Appearance<br>Bilirubin<br>Blood - Dip | |
| | | | | | Blood - Haemolysed / Non-Haemolysed<br>Colour<br>Glucose<br>Ketones<br>Leukocytes<br>Nitrite<br>Protein<br>Specific Gravity<br>Urobilinogen<br>pH | |
| | | | | | Interpretation<br>Sent for Microscopy<br>Comments | |

<sup>[1]</sup> NCS = Not clinically significant, CS = Clinically significant.

Programming note: The physician interpretation and microscopy (Yes/No) will be shown as an additional row at the end of each assessment, with the interpretation/microscopy outcome shown in the result column.

Programming note: for Blood parameter there is a Haemolysed/Non-Haemolysed as well as a result.

Version 01-00, 20DEC2022

# Listing 16.2.9. Urinalysis (TDL): Microscopy

| Treatment<br>Group | Participant | Visit | Sample Collection<br>Date / Time<br>(Study Day) | Urine<br>RBC | Urine<br>WBC | Cellular<br>casts | Granular<br>casts | Hyaline<br>casts | Urine<br>culture |
|---|---|---|---|---|---|---|---|---|---|
| xxxxxx | xxxxxx | xxxx | ddmmyyyy / hh:mm (xx) | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxx | xxxxxxxx |

ND = Not Done, A = Abnormal

Listing 16.2.10 Vital Signs

| Treatment<br>Group | Participant | Visit | Date | Assessment | Time Started<br>Supine | Collection<br>Time | Parameter | Result [1] | Change from<br>Baseline | Units | Comments |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1.1 | 1 / 0 / 2 | | 1.1 | 0 1 1 2 | | | | |
| XXXXXX | XXXXXX | XXXX | ddmmyyyy | 1 / 2 / 3 | hh:mm | hh:mm | Systolic BP | XXX | XXX | mmHg | |
| | | | | | | | Diastolic BP | XX | XX | mmHG | |
| | | | | | | | Heart Rate | XX | xx | bpm | |
| | | | | | | | Rep. Rate | XX | XX | breaths/min | |
| | | | | | | | SpO2 | xx | XX | % | |
| | | | | | | | Tympanic | | | | |
| | | | | | | | temperature | xx.x | xx.x | deg C | |
| | | | | | | | Interpretation | xxxxxxx | | | xxxxxx |

<sup>[1]</sup> NCS = Not clinically significant, CS = Clinically significant.\* = tympanic temperature >= 37.9 deg C.

Programming note: The physician interpretation will be shown as an additional row at the end of each assessment, with the interpretation outcome shown in the result column. Add  $\star$  to any temperature result >=37.9 deg C.

Listing 16.2.11 Spirometry

| Treatment | | | Date / Time | | | |
|---|---|---|---|---|---|---|
| Group | Participant | Visit | (Study Day) | Parameter | Result [1] | Units |
| XXXXXXX | xxxxxx | XXXX | Ddmmyyyy hh;mm (XX) | FEV1 (abs) | x.xx | L |
| | | | | FEV1 (% Pred) | xx | % |
| | | | | FEV1/FVC Ratio (abs) | xx | |
| | | | | FEV1/FVC Ratio (% Pred) | XX | % |
| | | | | FVC (abs) | x.xx | L |
| | | | | FVC (% Pred) | XX | % |
| | | | | FEV1 decreased by $> 15\%$ from baseline FEV1 or FVC $< 80\%$ of the predicted | Yes / No | |
| | | | | value? | Yes / No | |

Listing 16.2.12.1
Physical Examination

| Group | Participant | Visit | Date / Time<br>(Study Day) | Parameter | Finding | Comments |
|---|---|---|---|---|---|---|
| xxxxxx | XXXXX | XXXX | ddmmyyyy hh:mm<br>(Study Day) | General Appearance Eyes Ears Nose Throat Head and Neck Cranial Nerves/Nervous System Musculoskeletal Skin Cardiovascular Abdomen/GI System Respiratory System Chest - Auscultation Chest - Vocal Resonance Chest - Percussion Other Findings | Normal / Abnormal Not Clinically Significant / Abnormal Clinically Significant / Not Done | |

Listing 16.2.12.2
Rhinoscopic Examination

| Treatment D | | | Date / Time | Date / Time | | |
|---|---|---|---|---|---|---|
| Group | Participant | Visit | (Study Day) | Assessment | Level [1] | Comments |
| | | | ddmmyyyy hh:mm | | | |
| xxxxxxx | xxxxxx | xxxx | (Study Day) | Nasal Discharge - Left | | |
| | | | | Nasal Discharge - Right | | |
| | | | | Otitis - Left | | |
| | | | | Otitis - Right | | |
| | | | | Pharyngitis | | |
| | | | | Sinus Tenderness - Left | | |
| | | | | Sinus Tenderness - Right | | |
| | | | | New Wheezes, Rhonchi - Left | | |
| | | | | New Wheezes, Rhonchi - Right | | |

[1] Nasal Discharge: 0 = None, 1 = Clear, serous; scant but slightly increased, 2 = Clear to white, obvious increased volume, + / - minor blood streaks on tissue, 3 = Frankly prudent (yellow or green), or gross blood.

Otitis: NA = Tympanic membrane not visible, 0 = None, 1 = Dulled tympanic membrane, 2 = Inflamed, injected tympanic membrane, 3 = Retracted or bulging tympanic membrane, obvious air, fluid level.

Pharyngitis: 0 = None, 1 = Mild and / or patchy erythema, 2 = Marked and / or confluent erythema, 3 = Erythema and purulent exudate.

Sinus Tenderness: 0 = None, 1 = Mild tenderness, 2 = Moderate tenderness, 3 = Severe tenderness or overlying erythema.

New Wheezes, Rhonchi: 0 = None, 1 = Mild wheezes or rhonchi, 2 = Scattered wheezes or rhonchi, 3 = Widespread wheezes.

Listing 16.2.111 ECG

| Preatment<br>Group Pa | Participant | Visit | Date | Time Started in Resting Position | Time Performed | Parameter | Result [1] | Units | Comments |
|---|---|---|---|---|---|---|---|---|---|
| (XXXXX X) | xxxxx | XXXX | ddmmyyyy | hh:mm | hh:mm | HR PR QRS QT QTc QTcB QTcF RR | XXX XXX XXX XXX XXX XXX XXX Normal / Abnormal NCS / Abnormal CS | bpm<br>ms<br>ms<br>ms<br>ms<br>ms<br>ms<br>ms | xxxxxx |

<sup>[1]</sup> NCS = Not clinically significant, CS = Clinically significant.

Programming note: The physician interpretation will be shown as an additional row at the end of each assessment, with the interpretation outcome shown in the result column.

Listing 16.2.14 Visit Dates

| Treatment<br>Group | Participant | Visit | Date | Source of Unscheduled Visit Comments | Comments |
|---|---|---|---|---|---|
| xxxxxxx | xxxxx | xxxx | ddmmyyyy | xxxxxxxxx | xxxxxxxxxxx |

Programming note: Unscheduled visits and visit information will be taken from specific database modules and the "Reason for additional collection" will be placed in the comments column in this listing.

# 15. APPENDICES

# 15.1. Study VIR-CST-001 assay cut-offs and reporting

| | | Associated | Assay Reporting | | |
|---|---|---|---|---|---|
| Analysis | Assay | units | Result | Reported result | S-cubed assigned value |
| | | Log <sub>10</sub><br>PFU/mL | ALOQ | ALOQ | 6.34 |
| | RSV Viral Culture<br>assay<br>(plaque assay) | | Quantifiable Titre | Value | Use reported value |
| RSV titre | | | DETECTED | DETECTED | 1.00 |
| (Viral Load) | | | NOT DETECTED | NOT DETECTED | 0 |
| | | | INVALID | INVALID | Missing data point |
| | | | NOT TESTED | N/A | Missing data point |
| | qRT-PCR<br>(in saline matrix) | Log <sub>10</sub><br>Copies/mL | Quantifiable Titre | Value | Use reported value |
| | | | DETECTED | DETECTED | 1.69 |
| RSV titre<br>(Viral Load) | | | NOT DETECTED | NOT DETECTED | 0 |
| (Viral Loud) | | | INVALID | INVALID | Missing data point |
| | | | NOT TESTED | N/A | Missing data point |
| | RSV | None | Quantifiable Titre | Value | Use reported value |
| RSV | Neutralisation Assay (virus focus reduction | | >4209 | >4209 | 4209 |
| antibody | | | <156 | <156 | 78 |
| titre | | | NDA | NDA | 10 |
| | neutralisation | | INVALID | INVALID | Missing data point |
| | assay) | | NOT TESTED | N/A | Missing data point |

N/A = not applicable; NDA = no detectable antibody.